CLINICAL TRIAL: NCT01636778
Title: Non-randomised, Open Label, Multi-centre Phase II Study to Assess the Efficacy and Safety of SB-497115-GR in Thrombocytopenic Subjects With Chronic Hepatitis C and Compensated Liver Cirrhosis.
Brief Title: Japanese Phase II Study of SB-497115-GR in Hepatitis C Virus Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116101
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C, Chronic
Keywords: Thrombocytopenia; Hepatitis C, chronic
MeSH Terms: conditions — Hepatitis C, Chronic; Thrombocytopenia | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SB-497115-GR (Experimental): investigational product for thrombocytopenia
  Interventions: Drug: SB-497115-GR

INTERVENTIONS:
Drug: SB-497115-GR — TPO receptor agonist to increase platelet count

SUMMARY:
The purpose of this study is to assess the ability of SB-497115-GR to raise platelet counts in thrombocytopenic patients with hepatitis C virus (HCV) infection (platelet count <80,000 /μL, suggestive of compensated cirrhosis) to a level desirable to initiate antiviral therapy and to assess the ability of SB-497115-GR to maintain platelet counts at a level sufficient to minimise dose reductions of pegylated interferon (Peg-IFN) and ribavirin (RBV) therapy with the expectation that a lower rate of Peg-IFN dose reduction and omission will translate to a higher rate of sustained viral response.

ELIGIBILITY:
Inclusion Criteria:

Subject is able to understand and comply with protocol requirements and instructions and is likely to complete the study as planned, as well as provided a written consent.

* A subject age between ≥20 and <75 years at time of informed consent.
* A subject who applies to one of the following:

Female subject with non-childbearing potential [i.e., physiologically incapable of becoming pregnant, who: has had a hysterectomy, or had a bilateral oophorectomy (ovariectomy), or had a bilateral tubal ligation, or is post-menopausal for greater than one year].

Female subject with childbearing potential, has a negative urine or serum pregnancy test at screening and within the 24-hour period prior to the first dose of SB-497115-GR, and completely abstains from intercourse or agree to use two of the following acceptable methods of contraception for 14 days before exposure to SB-497115-GR, throughout the clinical trial, and for 24 weeks after completion or premature discontinuation from the study.

Intrauterine device or intrauterine system that meets the effectiveness criteria as stated in the product label.

Male partner sterilization prior to the female subject's entry into the study, and this male is the sole partner for that subject.

Double-barrier contraception (condom with spermicidal jelly, or diaphragm with spermicide).

Male subject with childbearing potential partner completely abstains from intercourse or agree to use condom and diaphragm with spermicide.

* Subjects who were diagnosed as hepatitis C or compensated liver cirrhosis (Child-Pugh class A) without hepatic encephalopathy, or ascites. If there is a clear cirrhosis, treatment should be given with care as there is a potential of progressing to liver failure.
* Subjects who, in the opinion of the investigator, are appropriate candidates for Peg-IFN and RBV combination therapy for 48 weeks.
* HCV positive by TaqMan test at screening.
* Subject who fulfil all the organ functions below.

Items Values Platelet <80,000 /μL Haemoglobin ≥12.0 g/dL* Absolute neutrophil count (ANC) ≥1500 /μL* Creatinine clearance >50 mL/minute Total bilirubin <2.0 mg/dL Albumin >3.0 g/dL Prothrombin time >60%

*If the investigators consider the values are sufficient to give Peg-IFN/RBV, then a subject can be enrolled upon consulting the Medical Monitor.

Exclusion Criteria:

* Subject who relapsed or did not respond after 48 weeks of Peg-IFN/RBV therapy had been given with sufficient dose previously.
* Subject with history of IFN (including Peg-IFN) therapy or Peg-IFN/RBV therapy, but could not been treated with optimal Peg-IFN/RBV therapy due to the reasons other than thrombocytopenia.
* Subject who received IFN therapy (including Peg-IFN), antiviral therapy (excluding oseltamivir phosphate, etc.), immuno-modulatory treatment, radiotherapy or phlebotomy within 3 months (90 days) prior to the first dose of SB-497115-GR.
* Treatment with an investigational drug within 30 days prior to the first dose of SB-497115-GR or 5 half-lives of that investigational drug (whichever is longer).
* Subject with decompensated liver disease.
* Chronic liver disease other than chronic hepatitis C (e.g., autoimmune hepatitis, alcohol-induced hepatitis, drug-induced hepatitis, etc.).
* Subject with idiopathic thrombocytopenic purpura or active autoimmune disease.
* Subject who have had a malignancy diagnosed and/or treated within the past 5 years.
* Subjects who require endoscopic treatment for varices or documented history of clinically significant bleeding from oesophageal or gastric varices.
* Any disease condition associated with active bleeding or requiring anticoagulation with heparin or warfarin.
* Subject with serious cardiac, cerebrovascular, chronic pulmonary disease or interstitial lung disease, or documented history of any of these diseases.
* Pre-existing cardiac disease (congestive heart failure in New York Heart Association Grade III/IV), or arrhythmias known to involve the risk of thromboembolic events (e.g. atrial fibrillation), or subjects with a QTcF >450 msec or if with bundle brunch block, QTcF >480 msec.
* Subject with depression, psychiatric disorder requiring treatment or suicidal ideation or suicide attempt history, or history of these.
* Subject with uncontrolled hypertension (≥160 mmHg systolic or ≥100 mmHg diastolic).
* Subject with diabetes mellitus that can not be controlled by treatment.
* Thyroid dysfunction not adequately controlled.
* Subjects with haemoglobinopathies.
* History or current condition of seizure disorder.
* Subject who was positive for Human Immunodeficiency Virus (HIV) antibody or Hepatitis B Virus (HBV) antigen.
* Subject with arterial or venous thrombosis history or evidence of portal vein thrombosis on abdominal imaging (e.g., by computerized tomography or magnetic resonance imaging) within 3 months.
* History of alcohol/drug abuse or dependence.
* History of platelet clumping that prevents reliable measurement of platelet counts.
* Subjects planning to have cataract surgery.
* History of major organ transplantation.
* Known hypersensitivity to SB-497115-GR ingredients, IFN (including Peg-IFN), nucleoside analogues or biological agents (i.e., vaccines).
* Pregnant or nursing women or a male subject with pregnant partner.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- Japan (14):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Wakayama

REFERENCES:
- [Derived] Kawaguchi T, Komori A, Fujisaki K, Nishiguchi S, Kato M, Takagi H, Tanaka Y, Notsumata K, Mita E, Nomura H, Shibatoge M, Takaguchi K, Hattori T, Sata M, Koike K. Eltrombopag enables initiation and completion of pegylated interferon/ribavirin therapy in Japanese HCV-infected patients with chronic liver disease and thrombocytopenia. Exp Ther Med. 2019 Jul;18(1):596-604. doi: 10.3892/etm.2019.7616. Epub 2019 May 24. PMID 31258695

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with chronic hepatitis C (CHC) or compensated liver cirrhosis, who cannot start polyethylene glycol (Peg)-interferon (IFN)/ribavirin (RBV) therapy due to thrombocytopenia (platelet count <80 giga (10^9) cells per liter (Gi/L).
Pre-assignment Details: The total study duration was a maximum of 88 weeks, which consisted of a Screening Period of less than or equal to 45 days, the Pre-Antiviral Treatment Period (Part 1) from 1 up to 9 weeks and the Antiviral Treatment Period (Part 2) of 48 weeks and Follow-up Period of 24 weeks.
Groups:
- Eltrombopag Dose Escalation: Part 1: Participants with an initial platelet count of <80 Gi/L, received eltrombopag at 12.5 milligrams (mg) once daily (QD) for 2 weeks. After 2 weeks, if the platelet count was <100 Gi/L, participants underwent dose escalation to 25 mg QD (up to 2 weeks). If platelet counts still remained <100 Gi/L, further dose escalations to 37.5 mg QD (up to 2 weeks) and 50 mg QD (up to a maximum of 3 weeks) were allowed. Participants who achieved platelet counts >=100 Gi/L during Part1 (maximum of up to 9 weeks) were eligible to enter the Antiviral Treatment Period (Part 2), whereas those who failed to reach platelet counts >=100 Gi/L were discontinued from eltrombopag and progressed to the Follow-up Period.
- Eltrombopag + Antiviral Therapy: Part 2: Participants completing Part 1 continued on the same dose of eltrombopag received in Part 1 (dose that effectively raised platelets to >=100 Gi/L) in combination with antiviral therapy (Peg-IFN alfa-2a/RBV or Peg-IFN alfa-2b/RBV) for a duration of 48 weeks. Dose adjustments of eltrombobag were permitted up to 50mg QD in order to maintain an appropriate platelet count.
- Eltrombopag + Antiviral Therapy: Follow-up Period After Part: Participants who completed therapy or had early termination in Part 2 had three post-treatment follow-up visits at 4 weeks, 12 weeks and 24 weeks after the end or withdrawal of study treatment.
Period: Pre-Antiviral Treatment Period (Part 1)
Arm/Group | Eltrombopag Dose Escalation: Part 1 | Eltrombopag + Antiviral Therapy: Part 2 | Eltrombopag + Antiviral Therapy: Follow-up Period After Part
Started | 45 | 0 | 0
Completed | 41 | 0 | 0
Not Completed | 4 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 0
Not completed — Protocol-Defined Stopping Criteria | 1 | 0 | 0
Period: Antiviral Treatment Period (Part 2)
Arm/Group | Eltrombopag Dose Escalation: Part 1 | Eltrombopag + Antiviral Therapy: Part 2 | Eltrombopag + Antiviral Therapy: Follow-up Period After Part
Started | 0 | 41 | 0
Completed | 0 | 31 | 0
Not Completed | 0 | 10 | 0
Not completed — Adverse Event | 0 | 7 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Physician Decision | 0 | 2 | 0
Period: Follow-up Period After Part 2
Arm/Group | Eltrombopag Dose Escalation: Part 1 | Eltrombopag + Antiviral Therapy: Part 2 | Eltrombopag + Antiviral Therapy: Follow-up Period After Part
Started | 0 | 0 | 41
Completed | 0 | 0 | 37
Not Completed | 0 | 0 | 4
Not completed — Other | 0 | 0 | 1
Not completed — Not entered FU period after withdrawal | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Arm/Group | Eltrombopag Dose Escalation: Part 1
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.8 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 15
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 45
Diagnosis [Number; unit: Participants]
  Chronic hepatitis C | 23
  Liver cirrosis | 22
HCV genotype [Number; unit: Participants]
  1a | 0
  1b | 33
  2a | 6
  2b | 5
  Others | 1
Child-Pugh Class [Number; unit: Participants] — The Child-Pugh (CP) score (ranging from 5 to 15, with 5 being mild and 15 being severe) is calculated based on total bilirubin, serum albumin, international normalized ratio, ascites, and hepatic encephalopathy, is used to assess the severity of liver disease. A CP score of 5-6 = Class A (mild); 7-9 = Class B (moderate); >9 = Class C (severe).
  Participants
    A (Score 5 - 6) | 44
    B (Score 7 - 9) | 1
    C (Score > 9) | 0
Number of Participants with or without previous IFN use [Number; unit: Participants]
  Naïve | 24
  Experienced | 21
Baseline alanine transaminase (ALT) [Mean (Standard Deviation); unit: IU/L] | 78.2 (47.82)
Baseline Hepatitis C Virus (HCV) RNA [Mean (Standard Deviation); unit: Log IU/mL] | 6.41 (0.706)
Baseline platelet counts [Number; unit: Participants]
  <50 Gi Platelets/L | 8
  >=50 Gi Platelets/L | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Whose Platelet Count Increased From a Baseline Count of < 80 Gi/L to a Count >=100 Gi/L During Part 1
Description: Participants were assessed for a shift from a baseline platelet count of <80 Gi/L to a count >=100 Gi/L during Part 1(up to 9 weeks). Platelet counts were measured by blood draw.
Time Frame: From Baseline up to Week 9 in Part 1
Population: Full Analysis Set 1 (FAS1) Population: all participants enrolled in Part 1.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag Dose Escalation: Part 1
Number analyzed (Participants) | 45
Participants | 43

2. Primary Outcome: Number of Participants Whose Platelet Counts Maintained at >=50 Gi/L During Part 2
Description: Participants were assessed for continuously maintaining platelet counts >=50 Gi/L during Part 2.
  Platelet counts were measured by blood draw.
Time Frame: From Antiviral Baseline to up to Week 48 in Part 2
Population: Full Analysis Set 2 (FAS2) Population: all participants enrolled in Part 2.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
Participants | 36
Statistical Analysis 1: Comparison: Eltrombopag + Antiviral Therapy: Part 2; Test type: Superiority or Other; Percentage = 88, 95% CI 2-sided [74 to 96]

3. Secondary Outcome: Median Platelet Count at the Indicated Time Points in Part 1
Description: Platelet counts were measured by blood draw
Time Frame: Baseline, Week1, 2, 3, 4, 5, 6, 7, 8, 9, Withdrawal in Part 1
Population: FAS1 Population.
Measure: Median (Full Range); unit: 10^9 Cells Per Liter (Gi/L)
Arm/Group | Eltrombopag Dose Escalation: Part 1
Number analyzed (Participants) | 45
10^9 Cells Per Liter (Gi/L)
  Baseline, n=45 | 63.0 [34 to 78]
  Week 1, n=43 | 74.0 [36 to 108]
  Week 2, n=36 | 100.0 [43 to 248]
  Week 3, n=17 | 97.0 [48 to 153]
  Week 4, n=9 | 104.0 [48 to 137]
  Week 5, n=4 | 87.0 [49 to 132]
  Week 6, n=3 | 83.0 [53 to 93]
  Week 7, n=3 | 97.0 [56 to 103]
  Week 8, n=2 | 79.0 [63 to 95]
  Week 9, n=1 | 100.0 [100 to 100]
  Withdrawal, n=4 | 96 [48 to 115]

4. Secondary Outcome: Time in Weeks to Achieve Platelet Count >= 100 Gi/L
Description: Participants were assessed for achieving platelet counts >=100 Gi/L during Part 1. Platelet counts were measured by blood draw.
Time Frame: From Baseline up to Week 9 in Part 1
Population: FAS1 Population: all participants enrolled in Part 1.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag Dose Escalation: Part 1
Number analyzed (Participants) | 43
Participants
  Within 2 Weeks | 11
  Within 4 Weeks | 25
  Within 6 Weeks | 5
  Within 8 Weeks | 1
  Within 9 Weeks | 0
  Greater than 9 Weeks | 1

5. Secondary Outcome: Median Platelet Count at the Indicated Time Points in Part 2
Description: Platelet counts were measured by blood draw
Time Frame: Antiviral Baseline, Week 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, Withdrawal in Part 2
Population: FAS2 Population.
Measure: Median (Full Range); unit: Gi/L
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
Gi/L
  Antiviral Baseline, n=41 | 114.0 [100 to 248]
  Week 1, n=40 | 106.5 [50 to 431]
  Week 2, n=40 | 118.0 [58 to 309]
  Week 4, n=37 | 89.0 [43 to 126]
  Week 6, n=36 | 86.0 [38 to 130]
  Week 8, n=36 | 79.5 [53 to 130]
  Week 12, n=36 | 80.5 [55 to 161]
  Week 16, n=36 | 79.5 [49 to 128]
  Week 20, n=36 | 75.5 [54 to 119]
  Week 24, n=36 | 76.5 [29 to 128]
  Week 28, n=34 | 75.0 [49 to 128]
  Week 32, n=34 | 73.0 [30 to 161]
  Week 36, n=34 | 76.0 [43 to 148]
  Week 40, n=33 | 80.0 [48 to 135]
  Week 44, n=31 | 79.0 [37 to 172]
  Week 48, n=31 | 82.0 [49 to 170]
  Withdrawal, n=10 | 102.0 [54 to 207]

6. Secondary Outcome: Median Platelet Count at the Indicated Time Points During Follow-up Period After Part 2
Description: Platelet counts were measured by blood draw at specified timepoints.
Time Frame: Follow-up (FU) Baseline, FU Week 4, FU Week 12 and and FU Week 24 after Part 2
Population: FAS2 Population. Participants with any antiviral drugs during follow-up period after Part 2 are excluded from this analysis.
Measure: Median (Full Range); unit: Gi/L
Groups:
- Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2: Participants who completed therapy or had early termination in Part 2 had three post-treatment follow-up visits at 4 weeks, 12 weeks and 24 weeks after the end or withdrawal of study treatment.
Arm/Group | Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2
Number analyzed (Participants) | 34
Gi/L
  FU Baseline, n=34 | 86.5 [36 to 184]
  FU Week 4, n=34 | 82.5 [43 to 645]
  FU Week 12, n=34 | 70.0 [37 to 154]
  FU Week 24, n=31 | 63.0 [41 to 145]

7. Secondary Outcome: Minimum Platelet Count on Antiviral Therapy
Description: Participants were assessed for platelet counts during antiviral therapy in Part 2.
  Platelet counts were measured by blood draw.
Time Frame: From Antiviral Baseline to up to Week 48 in Part 2
Population: FAS2 Population: all participants enrolled in Part 2.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
Participants
  <25 Gi/L | 0
  >=25 to <50 Gi/L | 5
  >=50 to <100 Gi/L | 34
  >=100 to <150 Gi/L | 2
  >=150 to <200 Gi/L | 0
  >=200 to <400 Gi/L | 0
  >= 400 Gi/L | 0

8. Secondary Outcome: Dose of Eltrombopag That Enabled Initiation of Antiviral Therapy
Description: Participants received eltrombopag at escalating dosages until a platelet count of >=100 Gi/L was achieved in Part 1. Platelet counts were measured by blood draw.
Time Frame: From Baseline up to Week 9 in Part 1
Population: FAS1 Population: all participants enrolled in Part 1.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag Dose Escalation: Part 1
Number analyzed (Participants) | 45
Participants
  Eltrombopag 0 mg | 1
  Eltrombopag 12.5 mg | 25
  Eltrombopag 25 mg | 13
  Eltrombopag 37.5 mg | 0
  Eltrombopag 50 mg | 2
  Did not initiate antiviral therapy | 4

9. Secondary Outcome: Number of Antiviral Therapy Dose Reductions in Part 2
Description: Number of reductions in Part 2 of either Peg-IFN or RBV. Participants were assigned a score equal to the number of times antiviral therapy was reduced (0=no dose reductions [DRs]; 1=one DR; 2=two DRs; 3=three DRs; >3=more than three DRs). Where possible, every effort was made to maintain the recommended dose of antiviral therapy. However, where dose modification of antiviral therapy was required due to safety concerns, it was performed by the Investigator as per the region-specific product labels of Peg-IFN and/or RBV.
Time Frame: From Antiviral Baseline up to Week 48 in Part 2
Population: FAS2 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
Participants
  0 DR | 8
  1 DR | 9
  2 DR | 10
  3 DR | 3
  4 DR | 2
  5 DR | 1
  7 DR | 3
  8 DR | 1
  10 DR | 2

10. Secondary Outcome: Number of Participants With the Indicated Levels of Peg-IFN Alpha-2a Therapy Dose Reductions in Part 2
Description: Participants were assigned a score equal to the number of times their Peg-IFN alpha-2a dose of antiviral therapy was reduced (0=no dose reductions [DRs]; 1=one DR; 2=two DRs; 3=three DRs; >3=more than three DRs). Where possible, every effort was made to maintain the recommended dose of antiviral therapy. However, where dose modification of antiviral therapy was required due to safety concerns, it was performed by the Investigator as per the region-specific product labels of Peg-IFN.
Time Frame: From Antiviral Baseline up to Week 48 in Part 2
Population: FAS2 Population. Only those particpants who met the criteria for antiviral therapy dose reduction of Peg-IFN alpha-2a were analyzed.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 16
Participants
  0 DR | 4
  1 DR | 6
  2 DR | 4
  3 DR | 1
  >3 DR | 1

11. Secondary Outcome: Number of Participants With the Indicated Levels of Peg-IFN Alpha-2b Therapy Dose Reductions in Part 2
Description: Participants were assigned a score equal to the number of times their Peg-IFN alpha-2b dose of antiviral therapy was reduced (0=no dose reductions [DRs]; 1=one DR; 2=two DRs; 3=three DRs; >3=more than three DRs). Where possible, every effort was made to maintain the recommended dose of antiviral therapy. However, where dose modification of antiviral therapy was required due to safety concerns, it was performed by the Investigator as per the region-specific product labels of Peg-IFN.
Time Frame: From Antiviral Baseline up to Week 48 in Part 2
Population: FAS2 Population. Only those particpants who met the criteria for antiviral therapy dose reduction of Peg-IFN alpha-2b were analyzed.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 25
Participants
  0 DR | 16
  1 DR | 2
  2 DR | 4
  3 DR | 0
  >3 DR | 3

12. Secondary Outcome: Number of Participants With the Indicated Levels of RBV Therapy Dose Reductions in Part 2
Description: Participants were assigned a score equal to the number of times their RBV dose of antiviral therapy was reduced (0=no DRs; 1=one DR; 2=two DRs; 3=three DRs; >3=more than three DRs). Where possible, every effort was made to maintain the recommended dose of antiviral therapy. However, where dose modification of antiviral therapy was required due to safety concerns, it was performed by the Investigator as per the region-specific product labels of RBV
Time Frame: From Antiviral Baseline up to Week 48 in Part 2
Population: FAS2 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
Participants
  0 DR | 14
  1 DR | 12
  2 DR | 9
  3 DR | 3
  >3 DR | 3

13. Secondary Outcome: Time to First Dose Reduction of Antiviral Therapy in Part 2
Description: Time to first dose reduction was calucated as the time period from the first dose to the first dose reduction.
Time Frame: From Antiviral Baseline up to Week 48 in Part 2
Population: FAS2 Population.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 45
weeks
  Peg-IFN alfa-2a dose reduction, n=12 | 9.44 (12.556)
  Peg-IFN alfa-2b dose reduction, n=9 | 6.22 (6.944)
  RBV dose reduction, n=27 | 9.16 (6.611)

14. Secondary Outcome: Number of Participants Who Discontinued Antiviral Therapy in Part 2
Description: Dosing discontinuation is defined as the occurrence of stopping the medication. Dosing discontinuation of Antviral Therapy was assessed up to 48 weeks in Part 2
Time Frame: From Antiviral Baseline up to Week 48 in Part 2
Population: FAS2 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
Participants | 8

15. Secondary Outcome: Number of Participants Who Discontinued Peg-IFN Alpha-2a Therapy in Part 2
Description: Dosing discontinuation is defined as the occurrence of stopping the medication. Dosing discontinuation of Peg-IFN alpha-2a therapy was assessed up to 48 weeks in Part 2
Time Frame: From Antiviral Baseline up to Week 48 in Part 2
Population: FAS2 Population. Only those particpants who received Peg-IFN alpha-2a antiviral therapy were analyzed.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 16
Participants | 1

16. Secondary Outcome: Number of Participants Who Discontinued Peg-IFN Alpha-2b Therapy in Part 2
Description: Dosing discontinuation is defined as the occurrence of stopping the medication. Dosing discontinuation of Peg-IFN alpha-2b therapy was assessed up to 48 weeks in Part 2
Time Frame: From Antiviral Baseline up to Week 48 in Part 2
Population: FAS2 Population. Only those particpants who received Peg-IFN alpha-2b antiviral therapy were analyzed.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 25
Participants | 7

17. Secondary Outcome: Number of Participants Achieving Adherence to Antiviral Therapy in Part 2
Description: Adherence to antiviral therapy was defined as receiving at least 80% of the prescribed dose (investigator prescribed) of Peg-IFN alfa and at least 80% of the prescribed dose (investigator prescribed) of RBV, for at least 80% of the planned duration
Time Frame: From Antiviral Baseline up to Week 48 in Part 2
Population: FAS2 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
Participants | 32

18. Secondary Outcome: Number of Participants Achieving Adherence to Peg-IFN Alpha 2a Antiviral Therapy in Part 2
Description: Adherence to antiviral therapy was defined as receiving at least 80% of the prescribed dose (investigator prescribed) of Peg-IFN alfa-2a and at least 80% of the prescribed dose (investigator prescribed) of RBV, for at least 80% of the planned duration.
Time Frame: From Antiviral Baseline up to Week 48 in Part 2
Population: FAS2 Population. Only those particpants who received Peg-IFN alpha-2a antiviral therapy were analyzed.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 16
Participants | 14

19. Secondary Outcome: Number of Participants Achieving Adherence to Peg-IFN Alpha-2b Antiviral Therapy in Part 2
Description: Adherence to antiviral therapy was defined as receiving at least 80% of the prescribed dose (investigator prescribed) of Peg-IFN alpha-2b and at least 80% of the prescribed dose (investigator prescribed) of RBV, for at least 80% of the planned duration.
Time Frame: From Antiviral Baseline up to Week 48 in Part 2
Population: FAS2 Population. Only those particpants who received Peg-IFN alpha-2b antiviral therapy were analyzed.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 25
Participants | 18

20. Secondary Outcome: Number of Participants With Sustained Virologic Response (SVR) in Part 2
Description: Participants with SVR were defined as those with undetectable Hepatitis C Virus (HCV) ribonucleic acid (RNA) at 24 weeks post-completion of treatment period Part 2
Time Frame: From Antiviral Baseline up to Week 48 in Part 2
Population: FAS2 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
Participants | 9

21. Secondary Outcome: Number of Participants With Rapid Virological Response (RVR) and Extended RVR (eRVR) in Part 2
Description: RVR is defined as the absence of detectable HCV RNA after 4 weeks of antiviral treatment. eRVR is defined as the absence of detectable HCV RNA between 4 weeks and 12 weeks after antiviral treatment.
Time Frame: From Antiviral Baseline up to Week 48 in Part 2
Population: FAS2 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
Participants
  RVR | 6
  eRVR | 5

22. Secondary Outcome: Number of Participants With Early Virological Response (EVR) and Complete EVR (cEVR) in Part 2
Description: EVR is defined as a clinically significant reduction from Baseline in HCV RNA (>=2 log10 decrease in HCV RNA or undetectable HCV RNA) after 12 weeks of antiviral treatment. cEVR, a subset of EVR, is defined exclusively as undetectable HCV RNA after 12 weeks of antiviral treatment.
Time Frame: From Antiviral Baseline up to Week 48 in Part 2
Population: FAS2 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
Participants
  EVR | 28
  cEVR | 18

23. Secondary Outcome: Number of Participants With End of Treatment Response (ETR) for Undetectable HCV RNA at the End of Peg-IFN/RBV Treatment in Part 2
Description: ETR is defined as undetectable HCV RNA at the end of Peg-IFN/RBV treatment.
Time Frame: From Antiviral Baseline up to Week 48 in Part 2
Population: FAS2 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
Participants | 19

24. Secondary Outcome: Mean Serum HCV RNA at the Indicated Time Points In Part 2
Description: The HCV is a small, enveloped, single-stranded, positive-sense RNA virus. Log-Transformed HCV RNA was assessed at Screening, Antiviral Baseline, Part 2 week 4, 12, 24, 36, 48 and at withdrawal.
Time Frame: Screening, Antviral baseline; Week 4, 12, 24, 36, 48, Withdrawal in Part 2
Population: FAS2 Population.
Measure: Mean (Standard Deviation); unit: Log international unit per milliliter
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
Log international unit per milliliter
  Screening, n=41 | 6.41 (0.726)
  Antiviral Baseline, n=41 | 6.37 (0.767)
  Week 4, n=37 | 3.77 (1.741)
  Week 12, n=36 | 2.52 (1.734)
  Week 24, n=36 | 2.46 (1.876)
  Week 36, n=34 | 2.69 (2.177)
  Week 48, n=31 | 2.63 (2.275)
  Withdrawal, n=10 | 3.87 (2.275)

25. Secondary Outcome: Mean Serum HCV RNA at the Indicated Time Points During Follow-up Period After Part 2
Description: The HCV is a small, enveloped, single-stranded, positive-sense RNA virus. Log-Transformed HCV RNA was assessed at FU Baseline, FU Week 12 and FU Week 24 during Follow-up Period after Part 2
Time Frame: FU Baseline, FU Week 12 and FU Week 24 after Part 2
Population: FAS2 Population. Participants with any antiviral drugs during follow-up period after Part 2 were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: Log international unit per milliliter
Arm/Group | Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2
Number analyzed (Participants) | 34
Log international unit per milliliter
  FU Baseline, n=34 | 3.10 (2.422)
  FU Week 12, n=34 | 5.04 (2.551)
  FU Week 24, n=31 | 4.82 (2.436)

26. Secondary Outcome: Number of Participants With Any Adverse Event (AE) and Any Serious Adverse Event (SAE) in Part1
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death; was life threatening; required hospitalization or prolongation of existing hospitalization; resulted in disability/incapacity; was a congenital anomaly/birth defect.
Time Frame: From Baseline up to week 9 in Part 1
Population: Safety Population 1 (SP1) : consisted of all participants who were enrolled in Part 1 and received at least one dose of eltrombopag.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag Dose Escalation: Part 1
Number analyzed (Participants) | 45
Participants
  Any AE | 13
  Any SAE | 0
  Fatal AE | 0
  Drug-related AE | 4
  AE leading to withdrawal | 0
  SAE leading to withdrawal | 0
  On-going AE at the endo of study/withdrawal | 1

27. Secondary Outcome: Number of Participants With Any AE and Any SAE in Part 2
Description: as for outcome 26
Time Frame: From Antiviral Baseline up to Week 48 in Part 2
Population: Safety Population 2 (SP2): consisted of all participants who were enrolled in Part 2 and received at least one dose of eltrombopag.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
Participants
  Any AE | 41
  Any SAE | 3
  Fatal AE | 0
  Drug-related AE | 41
  AE leading to withdrawal | 9
  SAE leading to withdrawal | 3
  On-going AE at the end of study/withdrawal | 34

28. Secondary Outcome: Number of Participants With Any AE and Any SAE During Follow-up Period After Part 2
Description: as for outcome 26
Time Frame: From FU Baseline up to FU Week 24 after Part 2
Population: SP2 Population
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2
Number analyzed (Participants) | 41
Participants
  Any AE | 25
  Any SAE | 4
  Fatal AE | 0
  Drug-related AE | 6
  AE leading to withdrawal | 0
  SAE leading to withdrawal | 0
  On-going AE at the end of study/withdrawal | 16

29. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at the Indicated Time Points in Part 1 With Follow-up Period
Description: Participant's blood pressure was measured at the indicated time points during the study. Systolic blood pressure is a measure of blood pressure while the heart is beating. Diastolic blood pressure is a measure of blood pressure while the heart is relaxed. Mean change from Baseline was calculated as the value at the indicated time points minus the value at Baseline
Time Frame: Baseline; Week 1, 2, 3, 4, 5, 6, 7, 8, 9, Withdrawal in Part 1 and FU Week 4, FU Week 12, and FU Week 24
Population: SP1
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Eltrombopag Dose Escalation: Part 1
Number analyzed (Participants) | 45
Millimeter of mercury (mmHg)
  SBP, Week 1, n=38 | 0.9 (9.86)
  SBP, Week 2, n=30 | -1.7 (12.42)
  SBP, Week 3, n=11 | 2.8 (11.07)
  SBP, Week 4, n=6 | -2.8 (9.79)
  SBP, Week 5, n=3 | -1.0 (9.54)
  SBP, Week 6, n=3 | -4.0 (3.00)
  SBP, Week 7, n=3 | -1.3 (5.69)
  SBP, Week 8, n=2 | 12.0 (15.56)
  SBP, Week 9, n=1 | 3.0 (NA) — Forty subjects in Part1 achieved platelet counts >=100 Gi/L until Week 7 and progressed to Part2. Four subjects were withdrawn before Week 9. The number of subject at Week 9 in Part 1 was one; therefore the SD cannot be calculated.
  SBP, Withdrawal, n=4 | 13.5 (13.96)
  SBP, Follow Up, week 4, n=3 | -1.0 (8.54)
  SBP, Follow Up, week 12, n=3 | 9.0 (8.89)
  SBP, Follow Up, week 24, n=3 | 2.7 (10.07)
  DBP, Week 1, n=38 | -0.5 (8.81)
  DBP, Week 2, n=30 | -2.1 (8.04)
  DBP, Week 3, n=11 | -1.6 (7.98)
  DBP, Week 4, n=6 | -1.7 (8.04)
  DBP, Week 5, n=3 | -7.3 (9.87)
  DBP, Week 6, n=3 | -3.3 (7.64)
  DBP, Week 7, n=3 | -9.0 (7.00)
  DBP, Week 8, n=2 | 6.0 (14.14)
  DBP, Week 9, n=1 | -10.0 (NA) — Forty subjects in Part1 achieved platelet counts >=100 Gi/L until Week 7 and progressed to Part2. Four subjects were withdrawn before Week 9. The number of subject at Week 9 in Part 1 was one; therefore the SD cannot be calculated.
  DBP, Withdrawal, n=4 | 5.8 (12.09)
  DBP, FU Week 4, n=3 | 0.3 (5.51)
  DBP, FU Week 12, n=3 | 4.0 (10.39)
  DBP, FU Week 24, n=3 | -0.3 (1.53)

30. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at the Indicated Time Points in Part 2
Description: as for outcome 29
Time Frame: Baseline; Antiviral Baseline,Week 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, Withdrawal in Part 2
Population: SP2: consisted of all participants who were enrolled in Part 2 and received at least one dose of eltrombopag.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
mmHg
  SBP, Antiviral Baseline, n=40 | 0.2 (13.99)
  SBP, Week 1, n=40 | -5.9 (10.37)
  SBP, Week 2, n=40 | -8.7 (13.35)
  SBP, Week 4, n=37 | -5.2 (13.69)
  SBP, Week 6, n=36 | -3.9 (13.09)
  SBP, Week 8, n=36 | -6.0 (14.53)
  SBP, Week 12, n=36 | -5.7 (13.08)
  SBP, Week 16, n=36 | -5.5 (16.52)
  SBP, Week 20, n=36 | -4.4 (15.18)
  SBP, Week 24, n=36 | -2.1 (15.70)
  SBP, Week 28, n=34 | -6.3 (15.76)
  SBP, Week 32, n=34 | -5.2 (17.60)
  SBP, Week 36, n=34 | -5.6 (15.36)
  SBP, Week 40, n=33 | -5.1 (13.47)
  SBP, Week 44, n=31 | -4.6 (16.60)
  SBP, Week 48, n=31 | -2.9 (12.37)
  SBP, withdrawal, n=10 | 0.5 (17.26)
  DBP, Antiviral Baseline, n=40 | -0.4 (6.35)
  DBP, Week 1, n=40 | -3.5 (9.28)
  DBP, Week 2, n=40 | -4.0 (9.59)
  DBP, Week 4, n=37 | -3.5 (9.81)
  DBP, Week 6, n=36 | -3.9 (9.16)
  DBP, Week 8, n=36 | -6.0 (9.62)
  DBP, Week 12, n=36 | -5.9 (10.07)
  DBP, Week 16, n=36 | -4.7 (9.94)
  DBP, Week 20, n=36 | -5.7 (11.17)
  DBP, Week 24, n=36 | -4.5 (12.34)
  DBP, Week 28, n=34 | -7.9 (11.48)
  DBP, Week 32, n=34 | -7.1 (11.97)
  DBP, Week 36, n=34 | -5.4 (9.96)
  DBP, Week 40, n=33 | -6.8 (9.69)
  DBP, Week 44, n=31 | -5.8 (12.18)
  DBP, Week 48, n=31 | -3.8 (8.36)
  DBP, withdrawal, n=10 | -2.4 (8.24)

31. Secondary Outcome: Mean Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at the Indicated Time Points During Follow-up Period After Part 2
Description: Participant's blood pressure was measured at the indicated time points during the study. Systolic blood pressure is a measure of blood pressure while the heart is beating. Diastolic blood pressure is a measure of blood pressure while the heart is relaxed.
Time Frame: FU Baseline, FU Week 4, FU Week 12 and FU Week 24 after Part 2
Population: SP2 Population.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2
Number analyzed (Participants) | 40
mmHg
  SBP, FU Baseline, n=40 | 126.5 (11.30)
  SBP, FU Week 4, n=40 | 125.4 (11.74)
  SBP, Week 12, n=40 | 126.7 (10.86)
  SBP, Week 24, n=37 | 128.4 (12.68)
  DBP, FU Baseline, n=40 | 73.8 (8.85)
  DBP, FU Week 4, n=40 | 74.3 (8.91)
  DBP, FU Week 12, n=40 | 76.2 (9.40)
  DBP, FU Week 24, n=37 | 75.7 (9.48)

32. Secondary Outcome: Mean Change From Baseline in Heart Rate at the Indicated Time Points in Part 1 With Follow-up Period
Description: The heart rate was measured in participants at the indicated time points. Mean change from Baseline was calculated as the value at the indicated time points minus the value at Baseline.
Time Frame: Baseline; Week 1, 2, 3, 4, 5, 6, 7, 8, 9, Withdrawal in Part 1 and FU Week 4, FU Week 12, FU Week 24
Population: SP1 Population.
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Eltrombopag Dose Escalation: Part 1
Number analyzed (Participants) | 45
Beats per minute (bpm)
  Week 1, n=38 | 0.1 (7.07)
  Week 2, n=30 | -0.1 (7.42)
  Week 3, n=11 | 0.1 (4.50)
  Week 4, n=6 | 2.8 (4.07)
  Week 5, n=3 | 0.3 (7.37)
  Week 6, n=3 | 2.0 (5.29)
  Week 7, n=3 | 3.0 (7.00)
  Week 8, n=2 | -1.0 (5.66)
  Week 9, n=1 | -4.0 (NA) — Forty subjects in Part1 achieved platelet counts >=100 Gi/L until Week 7 and progressed to Part2. Four subjects were withdrawn before Week 9. The number of subject at Week 9 in Part 1 was one; therefore the SD cannot be calculated.
  Withdrawal, n=4 | 2.8 (8.30)
  FU Week 4, n=3 | 0.7 (12.66)
  FU Week 12, n=3 | 3.7 (9.07)
  FU Week 24, n=3 | 2.0 (9.54)

33. Secondary Outcome: Mean Change From Antiviral Baseline in Heart Rate at the Indicated Time Points in Part 2
Description: The heart rate was measured in participants at the indicated time points. Mean change from Antiviral Baseline was calculated as the value at the indicated time points minus the value at Antiviral Baseline.
Time Frame: Antiviral Baseline, Week 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, Withdrawal in Part 2
Population: SP2 Population.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
bpm
  Antiviral Baseline, n=40 | 0.4 (7.56)
  Week 1, n=40 | -3.5 (9.51)
  Week 2, n=40 | 1.0 (9.57)
  Week 4, n=37 | 3.9 (9.29)
  Week 6, n=36 | 5.9 (9.78)
  Week 8, n=36 | 4.7 (10.60)
  Week 12, n=36 | 5.8 (10.34)
  Week 16, n=36 | 6.2 (9.91)
  Week 20, n=36 | 4.5 (10.54)
  Week 24, n=36 | 4.5 (9.79)
  Week 28, n=34 | 5.6 (9.85)
  Week 32, n=34 | 3.6 (8.80)
  Week 36, n=34 | 4.7 (9.07)
  Week 40, n=33 | 5.2 (8.20)
  Week 44, n=31 | 5.2 (7.11)
  Week 48, n=31 | 3.6 (7.18)
  Withdrawal, n=10 | 5.1 (11.86)

34. Secondary Outcome: Mean Heart Rate at the Indicated Time Points During Follow-up Period After Part 2
Description: The heart rate was measured in participants at the indicated time points.
Time Frame: FU Baseline, FU Week 4, FU Week 12 and FU Week 24 after Part 2
Population: SP2 Population.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2
Number analyzed (Participants) | 40
bpm
  FU Baseline, n=40 | 78.3 (8.77)
  FU Week 4, n=40 | 79.5 (9.38)
  FU Week 12, n=40 | 74.0 (8.64)
  FU Week 24, n=37 | 74.6 (9.58)

35. Secondary Outcome: Mean Change From Baseline in Weight at the Indicated Time Points in Part 1 With Follow-up Period
Description: The weight of participants was recorded at the indicated time points. Mean change from Baseline was calculated as the value at the indicated time points minus the value at Baseline.
Time Frame: Baseline; Week 1, 2, 3, 4, 5, 6, 7, 8, 9, Withdrawal in Part 1 and FU Week 4, FU Week 12, FU Week 24
Population: SP1 Population.
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Eltrombopag Dose Escalation: Part 1
Number analyzed (Participants) | 45
Kilogram (kg)
  Week 1, n=38 | 0.09 (0.807)
  Week 2, n=30 | 0.05 (1.239)
  Week 3, n=11 | 0.75 (1.196)
  Week 4, n=6 | 1.15 (0.931)
  Week 5, n=3 | 1.00 (1.400)
  Week 6, n=3 | 1.03 (0.723)
  Week 7, n=3 | 0.57 (1.159)
  Week 8, n=2 | 0.15 (1.909)
  Week 9, n=1 | 0.20 (NA) — Forty subjects in Part1 achieved platelet counts >=100 Gi/L until Week 7 and progressed to Part2. Four subjects were withdrawn before Week 9. The number of subject at Week 9 in Part 1 was one; therefore the SD cannot be calculated.
  Withdrawal, n=4 | 0.30 (1.519)
  FU Week 4, n=3 | 0.90 (1.212)
  FU Week 12, n=3 | 0.93 (3.009)
  FU Week 24, n=3 | 1.17 (2.894)

36. Secondary Outcome: Mean Change From Baseline in Weight at the Indicated Time Points in Part 2
Description: as for outcome 35
Time Frame: Baseline; Antiviral Baseline, Week 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, Withdrawal in Part 2
Population: SP2 Population.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
kg
  Antivital Baseline, n=40 | 0.04 (1.336)
  Week 1, n=40 | -0.95 (1.131)
  Week 2, n=40 | -1.14 (1.314)
  Week 4, n=37 | -1.04 (1.060)
  Week 6, n=36 | -1.05 (1.344)
  Week 8, n=36 | -1.28 (1.581)
  Week 12, n=36 | -1.73 (1.887)
  Week 16, n=36 | -2.13 (2.175)
  Week 20, n=36 | -2.49 (2.265)
  Week 24, n=36 | -3.11 (2.488)
  Week 28, n=34 | -3.00 (3.104)
  Week 32, n=34 | -3.16 (3.100)
  Week 36, n=34 | -3.43 (3.188)
  Week 40, n=33 | -3.61 (3.000)
  Week 44, n=31 | -3.39 (3.018)
  Week 48, n=31 | -3.76 (2.950)
  Withdrawal, n=10 | -3.04 (3.584)

37. Secondary Outcome: Mean Weight at the Indicated Time Points During Follow-up Period After Part 2
Description: The weight of participants was recorded at the indicated time points.
Time Frame: FU Baseline, FU Week 4, FU Week 12 and FU Week 24 after Part 2
Population: SP2 Population
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2
Number analyzed (Participants) | 40
kg
  FU Baseline, n=40 | 55.77 (11.403)
  FU Week 4, n=40 | 56.37 (11.627)
  FU Week 12, n=40 | 57.05 (11.841)
  FU Week 24, n=37 | 57.84 (12.478)

38. Secondary Outcome: Mean Change From Baseline in Body Temperature at the Indicated Time Points in Part 1 With Follow-up Period
Description: The Body temperature of participants was recorded at the indicated time points. Mean change from Baseline was calculated as the value at the indicated time points minus the value at Baseline.
Time Frame: Baseline; Week 1, 2, 3, 4, 5, 6, 7, 8, 9, Withdrawal in Part 1 and FU Week 4, FU Week 12, FU Week 24
Population: SP1 Population.
Measure: Mean (Standard Deviation); unit: Degrees centigrade
Arm/Group | Eltrombopag Dose Escalation: Part 1
Number analyzed (Participants) | 45
Degrees centigrade
  Week 1, n=38 | -0.04 (0.439)
  Week 2, n=30 | 0.03 (0.445)
  Week 3, n=11 | 0.06 (0.284)
  Week 4, n=6 | 0.07 (0.367)
  Week 5, n=3 | -0.07 (0.153)
  Week 6, n=3 | -0.10 (0.173)
  Week 7, n=3 | -0.40 (0.100)
  Week 8, n=2 | -0.50 (0.141)
  Week 9, n=1 | -1.10 (NA) — Forty subjects in Part1 achieved platelet counts >=100 Gi/L until Week 7 and progressed to Part2. Four subjects were withdrawn before Week 9. The number of subject at Week 9 in Part 1 was one; therefore the SD cannot be calculated.
  Withdrawal, n=4 | -0.18 (0.171)
  FU Week 4, n=3 | 0.07 (0.153)
  FU Week 12, n=3 | -0.23 (0.493)
  FU Week 24, n=3 | -0.17 (0.306)

39. Secondary Outcome: Mean Change From Baseline in Body Temperature at the Indicated Time Points in Part 2
Description: as for outcome 38
Time Frame: Baseline; Antiviral Baseline,Week 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, Withdrawal in Part 2
Population: SP2 Population.
Measure: Mean (Standard Deviation); unit: Degrees centigrade
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
Degrees centigrade
  Antiviral Baseline, n=41 | 0.08 (0.662)
  Week 1, n=40 | 0.09 (0.398)
  Week 2, n=40 | 0.17 (0.459)
  Week 4, n=37 | 0.16 (0.439)
  Week 6, n=36 | 0.19 (0.499)
  Week 8, n=36 | 0.22 (0.426)
  Week 12, n=36 | 0.28 (0.440)
  Week 16, n=36 | 0.22 (0.392)
  Week 20, n=36 | 0.20 (0.386)
  Week 24, n=36 | 0.26 (0.422)
  Week 28, n=34 | 0.27 (0.424)
  Week 32, n=34 | 0.21 (0.435)
  Week 36, n=34 | 0.22 (0.462)
  Week 40, n=33 | 0.26 (0.374)
  Week 44, n=31 | 0.20 (0.492)
  Week 48, n=31 | 0.15 (0.498)
  Withdrawal, n=10 | 0.38 (0.724)

40. Secondary Outcome: Mean Body Temperature at the Indicated Time Points During Follow-up Period After Part 2
Description: The Body temperature of participants was recorded at the indicated time points..
Time Frame: FU Baseline, FU Week 4, FU Week 12 and FU Week 24 after Part 2
Population: SP2 Population
Measure: Mean (Standard Deviation); unit: Degrees centigrade
Arm/Group | Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2
Number analyzed (Participants) | 40
Degrees centigrade
  FU Baseline, n=40 | 36.44 (0.417)
  FU Week 4, n=40 | 36.37 (0.360)
  FU Week 12, n=40 | 36.29 (0.350)
  FU Week 24, n=37 | 36.90 (0.377)

41. Secondary Outcome: Mean Change From Baseline in Body Mass Index (BMI) at the Indicated Time Points in Part 1 With Follow-up Periodc
Description: The BMI for participants was calculated at the indicated time points as body weight in kilograms divided by height in meters squared. Mean change from Baseline was calculated as the value at the indicated time points minus the value at Baseline
Time Frame: Baseline; Week 1, 2, 3, 4, 5, 6, 7, 8, 9, Withdrawal in Part 1 and FU Week 4, FU Week 12, FU Week 24
Population: SP1 Population.
Measure: Mean (Standard Deviation); unit: kilogram per meters squared (kg/m^2)
Arm/Group | Eltrombopag Dose Escalation: Part 1
Number analyzed (Participants) | 45
kilogram per meters squared (kg/m^2)
  Week 1, n=38 | 0.03 (0.302)
  Week 2, n=30 | 0.02 (0.457)
  Week 3, n=11 | 0.26 (0.415)
  Week 4, n=6 | 0.39 (0.325)
  Week 5, n=3 | 0.36 (0.504)
  Week 6, n=3 | 0.36 (0.248)
  Week 7, n=3 | 0.20 (0.417)
  Week 8, n=2 | 0.04 (0.704)
  Week 9, n=1 | 0.08 (NA) — Forty subjects in Part1 achieved platelet counts >=100 Gi/L until Week 7 and progressed to Part2. Four subjects were withdrawn before Week 9. The number of subject at Week 9 in Part 1 was one; therefore the SD cannot be calculated.
  Withdrawal, n=4 | 0.09 (0.572)
  FU, Week 4, n=3 | 0.34 (0.432)
  FU, Week 12, n=3 | 0.36 (1.084)
  FU, Week 24, n=3 | 0.41 (1.042)

42. Secondary Outcome: Mean Change From Baseline in BMI at the Indicated Time Points in Part 2
Description: as for outcome 41
Time Frame: Baseline; Antiviral Baseline,Week 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, Withdrawal in Part 2
Population: SP2 Population.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
kg/m^2
  Antiviral Baseline, n=40 | 0.01 (0.476)
  Week 1, n=40 | -0.37 (0.408)
  Week 2, n=40 | -0.44 (0.495)
  Week 4, n=37 | -0.41 (0.424)
  Week 6, n=36 | -0.42 (0.534)
  Week 8, n=36 | -0.51 (0.624)
  Week 12, n=36 | -0.70 (0.723)
  Week 16, n=36 | -0.86 (0.844)
  Week 20, n=36 | -1.01 (0.891)
  Week 24, n=36 | -1.25 (0.965)
  Week 28, n=34 | -1.21 (1.212)
  Week 32, n=34 | -1.28 (1.228)
  Week 36, n=34 | -1.38 (1.264)
  Week 40, n=33 | -1.45 (1.200)
  Week 44, n=31 | -1.36 (1.174)
  Week 48, n=31 | -1.50 (1.146)
  Withdrawal, n=10 | -1.23 (1.529)

43. Secondary Outcome: Mean BMI at the Indicated Time Points During Follow-up Period After Part 2
Description: The BMI for participants was calculated at the indicated time points as body weight in kilograms divided by height in meters squared.
Time Frame: FU Baseline, FU Week 4, FU Week 12 and FU Week 24 after Part 2
Population: SP2 Population
Measure: Mean (Standard Deviation); unit: kilogram per meters squared (kg/m^2)
Arm/Group | Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2
Number analyzed (Participants) | 40
kilogram per meters squared (kg/m^2)
  FU Baseline, n=40 | 21.89 (3.486)
  FU Week 4, n=40 | 22.11 (3.474)
  FU Week 12, n=40 | 22.37 (3.531)
  FU Week 24, n=37 | 22.54 (3.521)

44. Secondary Outcome: Number of Participants With the Indicated Shift From Baseline in Severity Grades for Clinical Chemistry Parameters Per Division of Acquired Immunodeficiency Syndrome (DAIDS) in Part 1
Description: Blood samples for the assessment of clinical chemistry parameters were taken at intervals in Part 1. Clinical chemistry parameters included albumin, alkaline phosphatase (ALP), ALT, aspartate amino transferase (AST), total bilirubin, calcium, creatinine, potassium, sodium, and uric acid. Per DAIDS toxicity table, the grade ranges for each parameter are as follows: Grade (G) 0=none, 1=mild; G2=moderate; G3=severe; G4=potentially life-threatening.
Time Frame: From Baseline up to Week 9
Population: SP1 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag Dose Escalation: Part 1
Number analyzed (Participants) | 45
Participants
  Albumin: Any Grade Increase | 5
  Albumin: Increase to G1 | 5
  Albumin: Increase to G2 | 0
  Albumin: Increase to G3 | 0
  Albumin: Increase to G4 | 0
  ALP: Any Grade Increase | 4
  ALP: Increase to G1 | 2
  ALP: Increase to G2 | 2
  ALP: Increase to G3 | 0
  ALP: Increase to G4 | 0
  ALT: Any Grade Increase | 5
  ALT: Increase to G1 | 1
  ALT: Increase to G2 | 2
  ALT: Increase to G3 | 2
  ALT: Increase to G4 | 0
  AST:Any Grade Increase | 9
  AST:Increase to G1 | 2
  AST:Increase to G2 | 5
  AST:Increase to G3 | 2
  AST:Increase to G4 | 0
  Total Bilirubin:Any Grade Increase | 8
  Total Bilirubin:Increase to G1 | 6
  Total Bilirubin:Increase to G2 | 2
  Total Bilirubin:Increase to G3 | 0
  Total Bilirubin:Increase to G4 | 0
  Calcium:Any Grade Increase | 5
  Calcium:Increase to G1 | 5
  Calcium:Increase to G2 | 0
  Calcium:Increase to G3 | 0
  Calcium:Increase to G4 | 0
  Creatinine:Any Grade Increase | 1
  Creatinine:Increase to G1 | 1
  Creatinine:Increase to G2 | 0
  Creatinine:Increase to G3 | 0
  Creatinine:Increase to G4 | 0
  Potassium:Any Grade Increase | 3
  Potassium:Increase to G1 | 3
  Potassium:Increase to G2 | 0
  Potassium:Increase to G3 | 0
  Potassium:Increase to G4 | 0
  Sodium:Any Grade Increase | 2
  Sodium:Increase to G1 | 2
  Sodium:Increase to G2 | 0
  Sodium:Increase to G3 | 0
  Sodium:Increase to G4 | 0
  Uric Acid:Any Grade Increase | 6
  Uric acid:Increase to G1 | 5
  Uric acid:Increase to G2 | 1
  Uric acid:Increase to G3 | 0
  Uric acid:Increase to G4 | 0

45. Secondary Outcome: Number of Participants With the Indicated Shift From Baseline in Severity Grades for Clinical Chemistry Parameters Per DAIDS in Part 2
Description: Blood samples for the assessment of clinical chemistry parameters were taken at intervals in Part 2. Clinical chemistry parameters included albumin, ALP, ALT, AST, total bilirubin, calcium, creatinine, potassium, sodium, and uric acid. Per DAIDS toxicity table, the grade ranges for each parameter are as follows: Grade (G) 0=none, 1=mild; G2=moderate; G3=severe; G4=potentially life-threatening.
Time Frame: From Antiviral Baseline up to Week 48
Population: SP2 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
Participants
  Albumin:Any Grade Increase | 18
  Albumin:Increase to G1 | 15
  Albumin:Increase to G2 | 3
  Albumin:Increase to G3 | 0
  Albumin:Increase to G4 | 0
  ALP:Any Grade Increase | 3
  ALP:Increase to G1 | 3
  ALP:Increase to G2 | 0
  ALP:Increase to G3 | 0
  ALP:Increase to G4 | 0
  ALT:Any Grade Increase | 14
  ALT:Increase to G1 | 1
  ALT:Increase to G2 | 6
  ALT:Increase to G3 | 6
  ALT:Increase to G4 | 1
  AST:Any Grade Increase | 22
  AST:Increase to G1 | 4
  AST:Increase to G2 | 11
  AST:Increase to G3 | 6
  AST:Increase to G4 | 1
  Total Bilirubin:Any Grade Increase | 20
  Total Bilirubin:Increase to G1 | 7
  Total Bilirubin:Increase to G2 | 9
  Total Bilirubin:Increase to G3 | 3
  Total Bilirubin:Increase to G4 | 1
  Calcium:Any Grade Increase | 31
  Calcium:Increase to G1 | 25
  Calcium:Increase to G2 | 6
  Calcium:Increase to G3 | 0
  Calcium:Increase to G4 | 0
  Creatinine:Any Grade Increase | 3
  Creatinine:Increase to G1 | 2
  Creatinine:Increase to G2 | 1
  Creatinine:Increase to G3 | 0
  Creatinine:Increase to G4 | 0
  Potassium:Any Grade Increase | 8
  Potassium:Increase to G1 | 8
  Potassium:Increase to G2 | 0
  Potassium:Increase to G3 | 0
  Potassium:Increase to G4 | 0
  Sodium:Any Grade Increase | 7
  Sodium:Increase to G1 | 7
  Sodium:Increase to G2 | 0
  Sodium:Increase to G3 | 0
  Sodium:Increase to G4 | 0
  Uric acid:Any Grade Increase | 13
  Uric acid:Increase to G1 | 9
  Uric acid:Increase to G2 | 4
  Uric acid:Increase to G3 | 0
  Uric acid:Increase to G4 | 0

46. Secondary Outcome: Number of Participants With the Indicated Shift From Baseline in Severity Grades for Clinical Chemistry Parameters Per DAIDS During Follow-up Period After Part 2
Description: as for outcome 45
Time Frame: From FU Week 4 to FU Week 24
Population: SP2 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2
Number analyzed (Participants) | 40
Participants
  Albumin:Any Grade Increase | 3
  Albumin:Increase to G1 | 2
  Albumin:Increase to G2 | 1
  Albumin:Increase to G3 | 0
  Albumin:Increase to G4 | 0
  ALP:Any Grade Increase | 5
  ALP:Increase to G1 | 4
  ALP:Increase to G2 | 1
  ALP:Increase to G3 | 0
  ALP:Increase to G4 | 0
  ALT:Any Grade Increase | 9
  ALT:Increase to G1 | 4
  ALT:Increase to G2 | 4
  ALT:Increase to G3 | 0
  ALT:Increase to G4 | 1
  AST:Any Grade Increase | 10
  AST:Increase to G1 | 3
  AST:Increase to G2 | 6
  AST:Increase to G3 | 0
  AST:Increase to G4 | 1
  Total Bilirubin:Any Grade Increase | 4
  Total Bilirubin:Increase to G1 | 2
  Total Bilirubin:Increase to G2 | 2
  Total Bilirubin:Increase to G3 | 0
  Total Bilirubin:Increase to G4 | 0
  Calcium:Any Grade Increase | 2
  Calcium:Increase to G1 | 2
  Calcium:Increase to G2 | 0
  Calcium:Increase to G3 | 0
  Calcium:Increase to G4 | 0
  Calcium serum high: Any Grade Increase | 0
  Calcium, serum high: Increase to G1 | 0
  Calcium, serum high: Increase to G2 | 0
  Calcium, serum high: Increase to G3 | 0
  Calcium, serum high: Increase to G4 | 0
  Calcium serum low: Any Grade Increase | 2
  Calcium, serum low: Increase to G1 | 2
  Calcium, serum low: Increase to G2 | 0
  Calcium, serum low: Increase to G3 | 0
  Calcium, serum low: Increase to G4 | 0
  Creatinine: Any Grade Increase | 1
  Creatinine: Increase to G1 | 1
  Creatinine: Increase to G2 | 0
  Creatinine: Increase to G3 | 0
  Creatinine: Increase to G4 | 0
  Potassium:Any Grade Increase | 3
  Potassium:Increase to G1 | 3
  Potassium:Increase to G2 | 0
  Potassium:Increase to G3 | 0
  Potassium:Increase to G4 | 0
  Potassium, serum high:Any Grade Increase | 0
  Potassium, serum high:Increase to G1 | 0
  Potassium, serum high:Increase to G2 | 0
  Potassium, serum high:Increase to G3 | 0
  Potassium, serum high:Increase to G4 | 0
  Potassium, serum low:Any Grade Increase | 3
  Potassium, serum low:Increase to G1 | 3
  Potassium, serum low:Increase to G2 | 0
  Potassium, serum low:Increase to G3 | 0
  Potassium, serum low:Increase to G4 | 0
  Sodium:Any Grade Increase | 1
  Sodium:Increase to G1 | 1
  Sodium:Increase to G2 | 0
  Sodium:Increase to G3 | 0
  Sodium:Increase to G4 | 0
  Sodium, serum high:Any Grade Increase | 1
  Sodium, serum high:Increase to G1 | 1
  Sodium, serum high:Increase to G2 | 0
  Sodium, serum high:Increase to G3 | 0
  Sodium, serum high:Increase to G4 | 0
  Sodium, serum low:Any Grade Increase | 0
  Sodium, serum low:Increase to G1 | 0
  Sodium, serum low:Increase to G2 | 0
  Sodium, serum low:Increase to G3 | 0
  Sodium, serum low:Increase to G4 | 0
  Uric acid:Any Grade Increase | 2
  Uric acid:Increase to G1 | 2
  Uric acid:Increase to G2 | 0
  Uric acid:Increase to G3 | 0
  Uric acid:Increase to G4 | 0

47. Secondary Outcome: Number of Participants With the Indicated Shifts From BL in Severity Grades for for Hematology Parameters Per DAIDS in Part 1
Description: Blood samples for the assessment of hematology parameters were taken at intervals throughout the study. Participants with the worst-case shift from BL in Part 1 are reported, per severity grades by DAIDS, for levels of hemoglobin (low=anemia), lymphocytes (low=lymphocytopenia), total neutrophils (low=neutropenia), and white blood cells (low=leukocytopenia). Per the DAIDS toxicity table, grade ranges for each parameter are as follows: Grade (G) 1=mild; G2=moderate; G3=severe; G4=potentially life-threatening.
Time Frame: From Baseline up to Week 9
Population: SP1 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag Dose Escalation: Part 1
Number analyzed (Participants) | 45
Participants
  Hemoglobin:Any Grade Increase | 1
  Hemoglobin:Increase to G1 | 1
  Hemoglobin:Increase to G2 | 0
  Hemoglobin:Increase to G3 | 0
  Hemoglobin:Increase to G4 | 0
  Lymphocytes:Any Grade Increase | 4
  Lymphocytes:Increase to G1 | 1
  Lymphocytes:Increase to G2 | 0
  Lymphocytes:Increase to G3 | 3
  Lymphocytes:Increase to G4 | 0
  Total Neutrophils:Any Grade Increase | 8
  Total Neutrophils:Increase to G1 | 6
  Total Neutrophils:Increase to G2 | 2
  Total Neutrophils:Increase to G3 | 0
  Total Neutrophils:Increase to G4 | 0
  Platelet count:Any Grade Increase | 0
  Platelet count:Increase to G1 | 0
  Platelet count:Increase to G2 | 0
  Platelet count:Increase to G3 | 0
  Platelet count:Increase to G4 | 0
  White Blood Cell count:Any Grade Increase | 7
  White Blood Cell count:Increase to G1 | 7
  White Blood Cell count:Increase to G2 | 0
  White Blood Cell count:Increase to G3 | 0
  White Blood Cell count:Increase to G4 | 0

48. Secondary Outcome: Number of Participants With the Indicated Shifts From BL in Severity Grades for for Hematology Parameters Per DAIDS in Part 2
Description: Blood samples for the assessment of hematology parameters were taken at intervals throughout the study. Participants with the worst-case shift from BL in Part 2 are reported, per severity grades by DAIDS, for levels of hemoglobin (low=anemia), lymphocytes (low=lymphocytopenia), total neutrophils (low=neutropenia), and white blood cells (low=leukocytopenia). Per the DAIDS toxicity table, grade ranges for each parameter are as follows: Grade (G) 1=mild; G2=moderate; G3=severe; G4=potentially life-threatening.
Time Frame: From Antiviral Baseline up to Week 48
Population: SP2 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
Participants
  Hemoglobin:Any Grade Increase | 38
  Hemoglobin:Increase to G1 | 3
  Hemoglobin:Increase to G2 | 11
  Hemoglobin:Increase to G3 | 24
  Hemoglobin:Increase to G4 | 0
  Lymphocytes:Any Grade Increase | 26
  Lymphocytes:Increase to G1 | 0
  Lymphocytes:Increase to G2 | 6
  Lymphocytes:Increase to G3 | 12
  Lymphocytes:Increase to G4 | 8
  Total Neutrophils:Any Grade Increase | 38
  Total Neutrophils:Increase to G1 | 8
  Total Neutrophils:Increase to G2 | 10
  Total Neutrophils:Increase to G3 | 16
  Total Neutrophils:Increase to G4 | 4
  Platelet count:Any Grade Increase | 5
  Platelet count:Increase to G1 | 0
  Platelet count:Increase to G2 | 0
  Platelet count:Increase to G3 | 5
  Platelet count:Increase to G4 | 0
  White Blood Cell count:Any Grade Increase | 38
  White Blood Cell count:Increase to G1 | 10
  White Blood Cell count:Increase to G2 | 18
  White Blood Cell count:Increase to G3 | 9
  White Blood Cell count:Increase to G4 | 1

49. Secondary Outcome: Number of Participants With the Indicated Shifts From BL in Severity Grades for Hematology Parameters Per DAIDS During Follow-up Period After Part 2
Description: as for outcome 48
Time Frame: From FU Week 4 to FU Week 24
Population: SP2 Population,
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2
Number analyzed (Participants) | 40
Participants
  Hemoglobin:Any Grade Increase | 2
  Hemoglobin:Increase to G1 | 2
  Hemoglobin:Increase to G2 | 0
  Hemoglobin:Increase to G3 | 0
  Hemoglobin:Increase to G4 | 0
  Lymphocytes:Any Grade Increase | 2
  Lymphocytes:Increase to G1 | 0
  Lymphocytes:Increase to G2 | 2
  Lymphocytes:Increase to G3 | 0
  Lymphocytes:Increase to G4 | 0
  Total Neutrophils:Any Grade Increase | 7
  Total Neutrophils:Increase to G1 | 3
  Total Neutrophils:Increase to G2 | 4
  Total Neutrophils:Increase to G3 | 0
  Total Neutrophils:Increase to G4 | 0
  Platelet count:Any Grade Increase | 15
  Platelet count:Increase to G1 | 0
  Platelet count:Increase to G2 | 8
  Platelet count:Increase to G3 | 7
  Platelet count:Increase to G4 | 0
  White Blood Cell count:Any Grade Increase | 6
  White Blood Cell count:Increase to G1 | 3
  White Blood Cell count:Increase to G2 | 3
  White Blood Cell count:Increase to G3 | 0
  White Blood Cell count:Increase to G4 | 0

50. Secondary Outcome: Number of Participants With the Indicated Urinalysis Parameters Tested by Dipstick at the Indicated Time Points in Part1 With Follow Up Period
Description: Urinalysis parameters included: urine bilirubin (UB), urine occult blood (UOB), urine glucose (UG), urine ketones (UK), pH, urine protein (UP), urine specific gravity (USG) and urine urobilinogen (UU). The dipstick test gives results in a semi-quantitative manner. UB was categorized as (-), negative (Neg). UOB was categorised as 1+, 2+, 3+, (-), Neg, trace. UG results were categorized as (-), 0.5, Neg. UK parameters were categorized as as (-), Neg. pH results were in the range of pH from 5-8.5 in increments of 0.5. UP was categorized as 1+, (-), Neg, trace. UU was categorized as 1+, 0.1, 1, 2, 4, Neg, trace, normal. USG results were in the range from 1.000-1.030 in increments of 0.001.
Time Frame: Screening, Baseline, Week 1, 2, 3, 4, 7, 8, Withdrawal, FU Week 24
Population: SP1 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag Dose Escalation: Part 1
Number analyzed (Participants) | 45
Participants
  Screening, UB, (-), n=45 | 6
  Screening, UB, Neg., n=45 | 39
  Screening, UOB, 1+, n=45 | 4
  Screening, UOB, 2+, n=45 | 1
  Screening, UOB, 3+, n=45 | 1
  Screening, UOB, (-), n=45 | 6
  Screening, UOB, Neg., n=45 | 31
  Screening, UOB, trace., n=45 | 2
  Screening, UG, (-), n=45 | 7
  Screening, UG, 0.5, n=45 | 1
  Screening, UG, Neg., n=45 | 37
  Screening, UK, (-), n=45 | 7
  Screening, UK, Neg., n=45 | 38
  Screening, pH, 5, n=45 | 1
  Screening, pH, 5.5, n=45 | 9
  Screening, pH, 6, n=45 | 9
  Screening, pH, 6.5, n=45 | 12
  Screening, pH, 7, n=45 | 9
  Screening, pH, 7.5, n=45 | 5
  Screening, UP, 1+., n=45 | 1
  Screening, UP, (-), n=45 | 5
  Screening, UP, Neg., n=45 | 35
  Screening, UP, trace, n=45 | 4
  Screening, UU, 1+, n=45 | 2
  Screening, UU, (-), n=45 | 1
  Screening, UU, 0.1, n=45 | 5
  Screening, UU, 1, n=45 | 6
  Screening, UU, 2, n=45 | 4
  Screening, UU, trace, n=45 | 19
  Screening, UU, normal, n=45 | 8
  Screening, USG, 1.005, n=45 | 2
  Screening, USG, 1.006, n=45 | 1
  Screening, USG, 1.007, n=45 | 2
  Screening, USG, 1.008, n=45 | 1
  Screening, USG, 1.009, n=45 | 1
  Screening, USG, 1.01, n=45 | 3
  Screening, USG, 1.011, n=45 | 2
  Screening, USG, 1.012, n=45 | 1
  Screening, USG, 1.013, n=45 | 1
  Screening, USG, 1.014, n=45 | 4
  Screening, USG, 1.015, n=45 | 4
  Screening, USG, 1.017, n=45 | 2
  Screening, USG, 1.018, n=45 | 4
  Screening, USG, 1.019, n=45 | 1
  Screening, USG, 1.02, n=45 | 8
  Screening, USG, 1.021, n=45 | 1
  Screening, USG, 1.022, n=45 | 1
  Screening, USG, 1.024, n=45 | 1
  Screening, USG, 1.025, n=45 | 1
  Screening, USG, 1.026, n=45 | 3
  Screening, USG, 1.03, n=45 | 1
  Baseline, UB, (-), n=45 | 6
  Baseline, UB, Neg., n=45 | 39
  Baseline, UOB, 1+, n=45 | 1
  Baseline, UOB, 2+, n=45 | 1
  Baseline, UOB, 3+, n=45 | 2
  Baseline, UOB, (-), n=45 | 6
  Baseline, UOB, Neg., n=45 | 32
  Baseline, UOB, trace., n=45 | 3
  Baseline, UG, 2+, n=45 | 1
  Baseline, UG, (-), n=45 | 7
  Baseline, UG, 0.1, n=45 | 1
  Baseline, UG, 0.5, n=45 | 1
  Baseline, UG, Neg., n=45 | 35
  Baseline, UK, (-), n=45 | 7
  Baseline, UK, Neg., n=45 | 38
  Baseline, pH, 5, n=45 | 2
  Baseline, pH, 5.5, n=45 | 8
  Baseline, pH, 6, n=45 | 13
  Baseline, pH, 6.5, n=45 | 11
  Baseline, pH, 7, n=45 | 7
  Baseline, pH, 7.5, n=45 | 3
  Baseline, pH, 8, n=45 | 1
  Baseline, UP, 1+., n=45 | 1
  Baseline, UP, (-), n=45 | 5
  Baseline, UP, Neg., n=45 | 36
  Baseline, UP, trace, n=45 | 3
  Baseline, UU, 1+, n=45 | 7
  Baseline, UU, (-), n=45 | 1
  Baseline, UU, 0.1, n=45 | 4
  Baseline, UU, 1, n=45 | 10
  Baseline, UU, 2, n=45 | 1
  Baseline, UU, trace, n=45 | 15
  Baseline, UU, normal, n=45 | 7
  Baseline, USG, 1.003, n=45 | 1
  Baseline, USG, 1.005, n=45 | 3
  Baseline, USG, 1.006, n=45 | 1
  Baseline, USG, 1.007, n=45 | 1
  Baseline, USG, 1.009, n=45 | 1
  Baseline, USG, 1.01, n=45 | 6
  Baseline, USG, 1.011, n=45 | 2
  Baseline, USG, 1.012, n=45 | 1
  Baseline, USG, 1.013, n=45 | 2
  Baseline, USG, 1.014, n=45 | 1
  Baseline, USG, 1.015, n=45 | 2
  Baseline, USG, 1.016, n=45 | 2
  Baseline, USG, 1.017, n=45 | 1
  Baseline, USG, 1.018, n=45 | 3
  Baseline, USG, 1.019, n=45 | 2
  Baseline, USG, 1.02, n=45 | 5
  Baseline, USG, 1.021, n=45 | 3
  Baseline, USG, 1.022, n=45 | 1
  Baseline, USG, 1.023, n=45 | 1
  Baseline, USG, 1.025, n=45 | 3
  Baseline, USG, 1.028, n=45 | 2
  Baseline, USG, 1.03, n=45 | 1
  Week 1, UB, Neg, n=1 | 1
  Week 1, UOB, Neg, n=1 | 1
  Week 1, UG, Neg, n=1 | 1
  Week 1, UK, Neg, n=1 | 1
  Week 1, pH, 7.5, n=1 | 1
  Week 1, UP, trace, n=1 | 1
  Week 1, USG, 1.021, n=1 | 1
  Week 1, UU, trace, n=1 | 1
  Week 2, UB, Neg, n=3 | 3
  Week 2, UOB, Neg, n=3 | 3
  Week 2, UG, 0.25, n=3 | 1
  Week 2, UG, Neg, n=3 | 2
  Week 2, UK, Neg, n=3 | 3
  Week 2, pH, 6, n=3 | 1
  Week 2, pH, 6.5, n=3 | 2
  Week 2, UP, Neg, n=3 | 3
  Week 2, USG, 1.016, Neg, n=3 | 1
  Week 2, USG, 1.019, n=3 | 1
  Week 2, USG, 1.02, n=3 | 1
  Week 2, UU, 0.1, n=3 | 1
  Week 2, UU, trace, n=3 | 1
  Week 2, UU, normal, n=3 | 1
  Week 3, UB, Neg, n=2 | 2
  Week 3, UOB, Neg, n=2 | 2
  Week 3, UG, >=1.0, n=2 | 1
  Week 3, UG, Neg, n=2 | 1
  Week 3, UK, Neg, n=2 | 2
  Week 3, pH, 6, n=2 | 1
  Week 3, pH, 6.5, n=2 | 1
  Week 3, UP, Neg, n=2 | 2
  Week 3, USG, 1.015, n=2 | 1
  Week 3, USG, 1.02, n=2 | 1
  Week 3, UU, 0.1, n=2 | 1
  Week 3, UU, 4, n=2 | 1
  Week 4, UB, Neg, n=5 | 5
  Week 4, UOB, Neg, n=5 | 5
  Week 4, UG, >=1.0, n=5 | 1
  Week 4, UG, Neg, n=5 | 4
  Week 4, UK, Neg, n=5 | 5
  Week 4, pH, 5.5, n=5 | 1
  Week 4, pH, 6, n=5 | 2
  Week 4, pH, 6.5, n=5 | 2
  Week 4, UP, Neg, n=5 | 5
  Week 4, USG, 1.015, n=5 | 1
  Week 4, USG, 1.02, n=5 | 2
  Week 4, USG, 1.025, n=5 | 1
  Week 4, USG, 1.026, n=5 | 1
  Week 4, UU, 1, n=5 | 2
  Week 4, UU, 2, n=5 | 1
  Week 4, UU, trace, n=5 | 2
  Week 7, UB, Neg, n=1 | 1
  Week 7, UOB, Neg, n=1 | 1
  Week 7, UG, 0.5, n=1 | 1
  Week 7, UK, Neg, n=1 | 1
  Week 7, pH, 7, n=1 | 1
  Week 7, UP, Neg, n=1 | 1
  Week 7, USG, 1.02, n=1 | 1
  Week 7, UU, 2, n=1 | 1
  Week 8, UB, Neg, n=2 | 2
  Week 8, UOB, Neg, n=2 | 1
  Week 8, UOB, trace, n=2 | 1
  Week 8, UG, 0.1 n=2 | 1
  Week 8, UG, Neg, n=2 | 1
  Week 8, UK, Neg, n=2 | 2
  Week 8, pH, 6, n=2 | 2
  Week 8, UP, Neg, n=2 | 2
  Week 8, USG, 1.023, n=2 | 1
  Week 8, USG, 1.025, n=2 | 1
  Week 8, UU, 0.1, n=2 | 1
  Week 8, UU, trace, n=2 | 1
  Withdrawal, UB, Neg, n=4 | 4
  Withdrawal, UOB, Neg, n=4 | 4
  Withdrawal, UG, 0.5, n=4 | 1
  Withdrawal, UG, Neg, n=4 | 3
  Withdrawal, UK, Neg, n=4 | 4
  Withdrawal, pH, 6, n=4 | 2
  Withdrawal, pH, 6.5, n=4 | 1
  Withdrawal, pH, 8, n=4 | 1
  Withdrawal, UP, Neg, n=4 | 4
  Withdrawal, USG, 1.008, n=4 | 1
  Withdrawal, USG, 1.01, n=4 | 1
  Withdrawal, USG, 1.018, n=4 | 1
  Withdrawal, USG, 1.025, n=4 | 1
  Withdrawal, UU, 1+, n=4 | 2
  Withdrawal, UU, 0.1, n=4 | 1
  Withdrawal, UU, 1, n=4 | 1
  FU, Week 24, UB, Neg, n=3 | 3
  FU Week 24, UOB, 1+, n=3 | 1
  FU Week 24, UOB, Neg, n=3 | 2
  FU Week 24, UG, Neg, n=3 | 3
  FU Week 24, UK, Neg, n=3 | 3
  FU Week 24, pH, 5.5, n=3 | 1
  FU Week 24, pH, 6, n=3 | 1
  FU Week 24, pH, 7, n=3 | 1
  FU Week 24, UP, Neg, n=3 | 3
  FU Week 24, USG, 1.004, n=3 | 1
  FU Week 24, USG, 1.01, n=3 | 1
  FU Week 24, USG, 1.02, n=3 | 1
  FU Week 24, UU, 0.1, n=3 | 1
  FU Week 24, UU, 1, n=3 | 1
  FU Week 24, UU, trace, n=3 | 1

51. Secondary Outcome: Number of Participants With the Indicated Urinalysis Parameters Tested by Dipstick at the Indicated Time Points in Part 2
Description: Urinalysis parameters included: UB, UOB, UG, UK, pH, UP, USG and UU. The dipstick test gives results in a semi-quantitative manner. UB was categorized as (-), negative (Neg). UOB was categorised as 1+, 2+, 3+, (-), Neg, trace. UG results were categorized as 1+, (-), 0.5, Neg. UK parameters were categorized as as (-), Neg. pH results were in the range of pH from 5-8.5 in increments of 0.5. UP was categorized as (-), Neg, trace. UU was categorized as 1+, 0.1, 1, 2, 4, Neg, trace, normal. USG results were in the range from 1.000-1.030 in increments of 0.001.
Time Frame: Antiviral Baseline,Week 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, Withdrawal
Population: SP2 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Part 2
Number analyzed (Participants) | 41
Participants
  Antiviral Baseline, UB, (-), n=41 | 5
  Antiviral Baseline, UB, Neg., n=41 | 36
  Antiviral Baseline, UOB, 1+, n=41 | 1
  Antiviral Baseline, UOB, (-), n=41 | 5
  Antiviral Baseline, UOB, Neg., n=41 | 33
  Antiviral Baseline, UOB, trace., n=41 | 2
  Antiviral Baseline, UG, 1+, n=41 | 1
  Antiviral Baseline, UG, 2+, n=41 | 1
  Antiviral Baseline, UG, (-), n=41 | 5
  Antiviral Baseline, UG, 0.25, n=41 | 1
  Antiviral Baseline, UG, 0.5, n=41 | 1
  Antiviral Baseline, UG, >=1.0, n=41 | 1
  Antiviral Baseline, UG, Neg., n=41 | 31
  Antiviral Baseline, UK, (-), n=41 | 5
  Antiviral Baseline, UK, Neg., n=41 | 35
  Antiviral Baseline, UK, trace, n=41 | 1
  Antiviral Baseline, pH, 5, n=41 | 1
  Antiviral Baseline, pH, 5.5, n=41 | 6
  Antiviral Baseline, pH, 6, n=41 | 11
  Antiviral Baseline, pH, 6.5, n=41 | 12
  Antiviral Baseline, pH, 7, n=41 | 6
  Antiviral Baseline, pH, 7.5, n=41 | 4
  Antiviral Baseline, pH, 8.5, n=41 | 1
  Antiviral Baseline, UP, (-), n=41 | 5
  Antiviral Baseline, UP, Neg, n=41 | 34
  Antiviral Baseline, UP, trace, n=41 | 2
  Antiviral Baseline, USG, 1.005, n=41 | 1
  Antiviral Baseline, USG, 1.006, n=41 | 1
  Antiviral Baseline, USG, 1.01, n=41 | 3
  Antiviral Baseline, USG, 1.011, n=41 | 4
  Antiviral Baseline, USG, 1.012, n=41 | 2
  Antiviral Baseline, USG, 1.013, n=41 | 2
  Antiviral Baseline, USG, 1.014, n=41 | 2
  Antiviral Baseline, USG, 1.015, n=41 | 4
  Antiviral Baseline, USG, 1.016, n=41 | 3
  Antiviral Baseline, USG, 1.017, n=41 | 1
  Antiviral Baseline, USG, 1.018, n=41 | 2
  Antiviral Baseline, USG, 1.019, n=41 | 1
  Antiviral Baseline, USG, 1.02, n=41 | 8
  Antiviral Baseline, USG, 1.021, n=41 | 1
  Antiviral Baseline, USG, 1.022, n=41 | 1
  Antiviral Baseline, USG, 1.023, n=41 | 1
  Antiviral Baseline, USG, 1.024, n=41 | 1
  Antiviral Baseline, USG, 1.025, n=41 | 1
  Antiviral Baseline, USG, 1.026, n=41 | 1
  Antiviral Baseline, USG, 1.027, n=41 | 1
  Antiviral Baseline, UU, 1+, n=41 | 3
  Antiviral Baseline, UU, 0.1, n=41 | 3
  Antiviral Baseline, UU, 1, n=41 | 6
  Antiviral Baseline, UU, 2, n=41 | 2
  Antiviral Baseline, UU, 4, n=41 | 2
  Antiviral Baseline, UU, Neg, n=41 | 1
  Antiviral Baseline, UU, trace, n=41 | 16
  Antiviral Baseline, UU, normal, n=41 | 8
  Week 4, UB, (-), n=37 | 6
  Week 4, UB, Neg, n=37 | 31
  Week 4, UOB, 2+, n=37 | 1
  Week 4, UOB, (-), n=37 | 6
  Week 4, UOB, Neg, n=37 | 30
  Week 4, UG, (-), n=37 | 6
  Week 4, UG, 0.1, n=37 | 1
  Week 4, UG, Neg, n=37 | 30
  Week 4, UK, (-), n=37 | 6
  Week 4, UK, Neg, n=37 | 31
  Week 4, pH, 5, n=37 | 1
  Week 4, pH, 5.5, n=37 | 4
  Week 4, pH, 6, n=37 | 9
  Week 4, pH, 6.5, n=37 | 12
  Week 4, pH, 7, n=37 | 6
  Week 4, pH, 7.5, n=37 | 4
  Week 4, pH, 8, n=37 | 1
  Week 4, UP, (-), n=37 | 4
  Week 4, UP, Neg, n=37 | 28
  Week 4, UP, trace, n=37 | 5
  Week 4, USG, 1.004, n=37 | 1
  Week 4, USG, 1.005, n=37 | 3
  Week 4, USG, 1.006, n=37 | 3
  Week 4, USG, 1.008, n=37 | 1
  Week 4, USG, 1.01, n=37 | 2
  Week 4, USG, 1.011, n=37 | 2
  Week 4, USG, 1.012, n=37 | 1
  Week 4, USG, 1.013, n=37 | 2
  Week 4, USG, 1.014, n=37 | 1
  Week 4, USG, 1.015, n=37 | 4
  Week 4, USG, 1.016, n=37 | 1
  Week 4, USG, 1.017, n=37 | 2
  Week 4, USG, 1.019, n=37 | 1
  Week 4, USG, 1.02, n=37 | 6
  Week 4, USG, 1.021, n=37 | 2
  Week 4, USG, 1.022, n=37 | 2
  Week 4, USG, 1.025, n=37 | 3
  Week 4, UU, 1+, n=37 | 3
  Week 4, UU, 0.1, n=37 | 2
  Week 4, UU, 1, n=37 | 7
  Week 4, UU, 2, n=37 | 2
  Week 4, UU, 4, n=37 | 1
  Week 4, UU, 8, n=37 | 1
  Week 4, UU, Neg, n=37 | 2
  Week 4, UU, trace, n=37 | 15
  Week 4, UU, normal, n=37 | 4
  Week 8, UB, (-), n=36 | 4
  Week 8, UB, 2, n=36 | 1
  Week 8, UB, Neg, n=36 | 31
  Week 8, UOB, 1+, n=36 | 1
  Week 8, UOB, 2+, n=36 | 1
  Week 8, UOB, (-), n=36 | 4
  Week 8, UOB, Neg, n=36 | 30
  Week 8, UG, 1+, n=36 | 1
  Week 8, UG, (-), n=36 | 5
  Week 8, UG, >=1.0, n=36 | 1
  Week 8, UG, Neg, n=36 | 29
  Week 8, UK, (-), n=36 | 5
  Week 8, UK, Neg, n=36 | 30
  Week 8, UK, trace, n=36 | 1
  Week 8, pH, 5, n=36 | 1
  Week 8, pH, 5.5, n=36 | 4
  Week 8, pH, 6, n=36 | 7
  Week 8, pH, 6.5, n=36 | 13
  Week 8, pH, 7, n=36 | 7
  Week 8, pH, 7.5, n=36 | 3
  Week 8, pH, 8, n=36 | 1
  Week 8, UP, 1+, n=36 | 2
  Week 8, UP, (-), n=36 | 2
  Week 8, UP, Neg, n=36 | 30
  Week 8, UP, trace, n=36 | 2
  Week 8, USG, 1.001, n=36 | 1
  Week 8, USG, 1.003, n=36 | 1
  Week 8, USG, 1.004, n=36 | 1
  Week 8, USG, 1.005, n=36 | 2
  Week 8, USG, 1.008, n=36 | 4
  Week 8, USG, 1.01, n=36 | 3
  Week 8, USG, 1.012, n=36 | 1
  Week 8, USG, 1.013, n=36 | 3
  Week 8, USG, 1.014, n=36 | 1
  Week 8, USG, 1.015, n=36 | 2
  Week 8, USG, 1.016, n=36 | 3
  Week 8, USG, 1.018, n=36 | 3
  Week 8, USG, 1.019, n=36 | 1
  Week 8, USG, 1.02, n=36 | 2
  Week 8, USG, 1.023, n=36 | 2
  Week 8, USG, 1.025, n=36 | 4
  Week 8, USG, <=1.005, n=36 | 1
  Week 8, USG, >=1.030, n=36 | 1
  Week 8, UU, 1+, n=36 | 5
  Week 8, UU, (-), n=36 | 1
  Week 8, UU, 0.1, n=36 | 2
  Week 8, UU, 1, n=36 | 7
  Week 8, UU, 2, n=36 | 1
  Week 8, UU, 4, n=36 | 3
  Week 8, UU, Neg, n=36 | 1
  Week 8, UU, trace, n=36 | 11
  Week 8, UU, normal, n=36 | 5
  Week 12, UB, (-), n=36 | 5
  Week 12, UB, Neg, n=36 | 31
  Week 12, UOB, (-), n=36 | 5
  Week 12, UOB, Neg, n=36 | 31
  Week 12, UG, (-), n=36 | 5
  Week 12, UG, 0.25, n=36 | 1
  Week 12, UG, Neg, n=36 | 30
  Week 12, UK, (-), n=36 | 5
  Week 12, UK, 0, n=36 | 1
  Week 12, UK, Neg, n=36 | 30
  Week 12, pH, 5, n=36 | 2
  Week 12, pH, 5.5, n=36 | 2
  Week 12, pH, 6, n=36 | 9
  Week 12, pH, 6.5, n=36 | 12
  Week 12, pH, 7, n=36 | 7
  Week 12, pH, 7.5, n=36 | 4
  Week 12, UP, 1+, n=36 | 2
  Week 12, UP, (-), n=36 | 3
  Week 12, UP, Neg, n=36 | 26
  Week 12, UP, trace, n=36 | 5
  Week 12, USG, 1.005, n=36 | 2
  Week 12, USG, 1.006, n=36 | 3
  Week 12, USG, 1.007, n=36 | 1
  Week 12, USG, 1.008, n=36 | 1
  Week 12, USG, 1.009, n=36 | 1
  Week 12, USG, 1.01, n=36 | 1
  Week 12, USG, 1.012, n=36 | 2
  Week 12, USG, 1.014, n=36 | 2
  Week 12, USG, 1.015, n=36 | 7
  Week 12, USG, 1.016, n=36 | 1
  Week 12, USG, 1.017, n=36 | 1
  Week 12, USG, 1.018, n=36 | 2
  Week 12, USG, 1.019, n=36 | 2
  Week 12, USG, 1.02, n=36 | 5
  Week 12, USG, 1.021, n=36 | 2
  Week 12, USG, 1.022, n=36 | 2
  Week 12, USG, 1.026, n=36 | 1
  Week 12, UU, 1+, n=36 | 1
  Week 12, UU, 0.1, n=36 | 3
  Week 12, UU, 1, n=36 | 4
  Week 12, UU, 2, n=36 | 3
  Week 12, UU, 4, n=36 | 2
  Week 12, UU, Neg, n=36 | 2
  Week 12, UU, trace, n=36 | 15
  Week 12, UU, normal, n=36 | 6
  Week 16, UB, (-), n=36 | 4
  Week 16, UB, Neg, n=36 | 32
  Week 16, UOB, 1+, n=36 | 2
  Week 16, UOB, 2+, n=36 | 2
  Week 16, UOB, 3+, n=36 | 1
  Week 16, UOB, (-), n=36 | 4
  Week 16, UOB, Neg, n=36 | 27
  Week 16, UG, (-), n=36 | 4
  Week 16, UG, 0.25, n=36 | 1
  Week 16, UG, Neg, n=36 | 31
  Week 16, UK, (-), n=36 | 4
  Week 16, UK, Neg, n=36 | 31
  Week 16, UK, trace, n=36 | 1
  Week 16, pH, 5, n=36 | 1
  Week 16, pH, 5.5, n=36 | 3
  Week 16, pH, 6, n=36 | 12
  Week 16, pH, 6.5, n=36 | 9
  Week 16, pH, 7, n=36 | 8
  Week 16, pH, 7.5, n=36 | 3
  Week 16, UP, 1+, n=36 | 1
  Week 16, UP, (-), n=36 | 3
  Week 16, UP, Neg, n=36 | 30
  Week 16, UP, trace, n=36 | 2
  Week 16, USG, 1.005, n=36 | 2
  Week 16, USG, 1.006, n=36 | 1
  Week 16, USG, 1.007, n=36 | 1
  Week 16, USG, 1.008, n=36 | 2
  Week 16, USG, 1.009, n=36 | 1
  Week 16, USG, 1.01, n=36 | 3
  Week 16, USG, 1.014, n=36 | 1
  Week 16, USG, 1.015, n=36 | 7
  Week 16, USG, 1.016, n=36 | 2
  Week 16, USG, 1.017, n=36 | 1
  Week 16, USG, 1.018, n=36 | 2
  Week 16, USG, 1.019, n=36 | 4
  Week 16, USG, 1.02, n=36 | 3
  Week 16, USG, 1.021, n=36 | 1
  Week 16, USG, 1.022, n=36 | 2
  Week 16, USG, 1.023, n=36 | 1
  Week 16, USG, 1.025, n=36 | 1
  Week 16, USG, 1.027, n=36 | 1
  Week 16, UU, 1+, n=36 | 5
  Week 16, UU, 2+, n=36 | 1
  Week 16, UU, 0.1, n=36 | 3
  Week 16, UU, 1, n=36 | 7
  Week 16, UU, 4, n=36 | 2
  Week 16, UU, Neg, n=36 | 3
  Week 16, UU, trace, n=36 | 11
  Week 16, UU, normal, n=36 | 4
  Week 20, UB, (-), n=36 | 2
  Week 20, UB, Neg, n=36 | 34
  Week 20, UOB, 1+, n=36 | 1
  Week 20, UOB, (-), n=36 | 2
  Week 20, UOB, Neg, n=36 | 33
  Week 20, UG, (-), n=36 | 2
  Week 20, UG, Neg, n=36 | 33
  Week 20, UG, trace, n=36 | 1
  Week 20, UK, (-), n=36 | 2
  Week 20, UK, Neg, n=36 | 34
  Week 20, pH, 5, n=36 | 4
  Week 20, pH, 5.5, n=36 | 1
  Week 20, pH, 6, n=36 | 10
  Week 20, pH, 6.5, n=36 | 8
  Week 20, pH, 7, n=36 | 6
  Week 20, pH, 7.5, n=36 | 7
  Week 20, UP, 1+, n=36 | 2
  Week 20, UP, (-), n=36 | 2
  Week 20, UP, Neg, n=36 | 30
  Week 20, UP, trace, n=36 | 2
  Week 20, USG, 1.004, n=36 | 1
  Week 20, USG, 1.005, n=36 | 2
  Week 20, USG, 1.006, n=36 | 1
  Week 20, USG, 1.007, n=36 | 2
  Week 20, USG, 1.009, n=36 | 3
  Week 20, USG, 1.01, n=36 | 3
  Week 20, USG, 1.013, n=36 | 3
  Week 20, USG, 1.014, n=36 | 2
  Week 20, USG, 1.015, n=36 | 2
  Week 20, USG, 1.016, n=36 | 2
  Week 20, USG, 1.017, n=36 | 2
  Week 20, USG, 1.018, n=36 | 3
  Week 20, USG, 1.019, n=36 | 1
  Week 20, USG, 1.02, n=36 | 2
  Week 20, USG, 1.021, n=36 | 2
  Week 20, USG, 1.025, n=36 | 3
  Week 20, USG, 1.029, n=36 | 1
  Week 20, USG, <=1.005, n=36 | 1
  Week 20, UU, 1+, n=36 | 3
  Week 20, UU, 2+, n=36 | 1
  Week 20, UU, 0.1, n=36 | 2
  Week 20, UU, 1, n=36 | 7
  Week 20, UU, 4, n=36 | 1
  Week 20, UU, 8, n=36 | 2
  Week 20, UU, Neg, n=36 | 2
  Week 20, UU, trace, n=36 | 13
  Week 20, UU, normal, n=36 | 5
  Week 24, UB, (-), n=36 | 2
  Week 24, UB, Neg, n=36 | 34
  Week 24, UOB, 1+, n=36 | 2
  Week 24, UOB, 3+, n=36 | 1
  Week 24, UOB, (-), n=36 | 2
  Week 24, UOB, Neg, n=36 | 30
  Week 24, UOB, trace, n=36 | 1
  Week 24, UG, (-), n=36 | 2
  Week 24, UG, 0.1, n=36 | 1
  Week 24, UG, Neg, n=36 | 33
  Week 24, UK, (-), n=36 | 2
  Week 24, UK, Neg, n=36 | 33
  Week 24, UK, trace, n=36 | 1
  Week 24, pH, 5, n=36 | 2
  Week 24, pH, 5.5, n=36 | 3
  Week 24, pH, 6, n=36 | 9
  Week 24, pH, 6.5, n=36 | 12
  Week 24, pH, 7, n=36 | 6
  Week 24, pH, 7.5, n=36 | 3
  Week 24, pH, 8.5, n=36 | 1
  Week 24, UP, (-), n=36 | 2
  Week 24, UP, Neg, n=36 | 28
  Week 24, UP, trace, n=36 | 6
  Week 24, USG, 1.008, n=36 | 1
  Week 24, USG, 1.009, n=36 | 3
  Week 24, USG, 1.01, n=36 | 3
  Week 24, USG, 1.011, n=36 | 4
  Week 24, USG, 1.012, n=36 | 2
  Week 24, USG, 1.013, n=36 | 1
  Week 24, USG, 1.014, n=36 | 2
  Week 24, USG, 1.015, n=36 | 7
  Week 24, USG, 1.016, n=36 | 1
  Week 24, USG, 1.017, n=36 | 1
  Week 24, USG, 1.018, n=36 | 1
  Week 24, USG, 1.019, n=36 | 2
  Week 24, USG, 1.021, n=36 | 2
  Week 24, USG, 1.022, n=36 | 1
  Week 24, USG, 1.023, n=36 | 1
  Week 24, USG, 1.025, n=36 | 2
  Week 24, USG, 1.03, n=36 | 1
  Week 24, USG, <=1.005, n=36 | 1
  Week 24, UU, 1+, n=36 | 2
  Week 24, UU, 3+, n=36 | 1
  Week 24, UU, 0.1, n=36 | 2
  Week 24, UU, 1, n=36 | 8
  Week 24, UU, 2, n=36 | 2
  Week 24, UU, 4, n=36 | 1
  Week 24, UU, Neg, n=36 | 2
  Week 24, UU, trace, n=36 | 13
  Week 24, UU, normal, n=36 | 5
  Week 28, UB, 1+, n=34 | 1
  Week 28, UB, (-), n=34 | 1
  Week 28, UB, Neg, n=34 | 32
  Week 28, UOB, 1+, n=34 | 1
  Week 28, UOB, (-), n=34 | 1
  Week 28, UOB, Neg, n=34 | 31
  Week 28, UOB, trace, n=34 | 1
  Week 28, UG, (-), n=34 | 1
  Week 28, UG, 0.5, n=34 | 1
  Week 28, UG, Neg, n=34 | 32
  Week 28, UK, (-), n=34 | 1
  Week 28, UK, Neg, n=34 | 32
  Week 28, UK, trace, n=34 | 1
  Week 28, pH, 5.5, n=34 | 1
  Week 28, pH, 6, n=34 | 12
  Week 28, pH, 6.5, n=34 | 11
  Week 28, pH, 7, n=34 | 6
  Week 28, pH, 7.5, n=34 | 3
  Week 28, pH, 8, n=34 | 1
  Week 28, UP, 1+, n=34 | 1
  Week 28, UP, Neg, n=34 | 27
  Week 28, UP, trace, n=34 | 6
  Week 28, USG, 1.005, n=34 | 3
  Week 28, USG, 1.007, n=34 | 2
  Week 28, USG, 1.008, n=34 | 1
  Week 28, USG, 1.009, n=34 | 2
  Week 28, USG, 1.011, n=34 | 1
  Week 28, USG, 1.012, n=34 | 2
  Week 28, USG, 1.013, n=34 | 1
  Week 28, USG, 1.015, n=34 | 2
  Week 28, USG, 1.016, n=34 | 1
  Week 28, USG, 1.017, n=34 | 2
  Week 28, USG, 1.018, n=34 | 1
  Week 28, USG, 1.019, n=34 | 2
  Week 28, USG, 1.02, n=34 | 3
  Week 28, USG, 1.022, n=34 | 1
  Week 28, USG, 1.023, n=34 | 2
  Week 28, USG, 1.024, n=34 | 2
  Week 28, USG, 1.025, n=34 | 4
  Week 28, USG, 1.027, n=34 | 1
  Week 28, USG, <=1.005, n=34 | 1
  Week 28, UU, 1+, n=34 | 4
  Week 28, UU, 0.1, n=34 | 3
  Week 28, UU, 1, n=34 | 6
  Week 28, UU, 2, n=34 | 2
  Week 28, UU, 4, n=34 | 3
  Week 28, UU, Neg, n=34 | 1
  Week 28, UU, trace, n=34 | 11
  Week 28, UU, normal, n=34 | 4
  Week 32, UB, (-), n=34 | 1
  Week 32, UB, Neg, n=34 | 33
  Week 32, UOB, 1+, n=34 | 1
  Week 32, UOB, (-), n=34 | 1
  Week 32, UOB, Neg, n=34 | 32
  Week 32, UG, (-), n=34 | 1
  Week 32, UG, Neg, n=34 | 33
  Week 32, UK, (-), n=34 | 1
  Week 32, UK, Neg, n=34 | 32
  Week 32, UK, trace, n=34 | 1
  Week 32, pH, 5, n=34 | 1
  Week 32, pH, 5.5, n=34 | 2
  Week 32, pH, 6, n=34 | 14
  Week 32, pH, 6.5, n=34 | 8
  Week 32, pH, 7, n=34 | 8
  Week 32, pH, 7.5, n=34 | 1
  Week 32, UP, (-), n=34 | 1
  Week 32, UP, Neg, n=34 | 29
  Week 32, UP, trace, n=34 | 4
  Week 32, USG, 1.005, n=34 | 2
  Week 32, USG, 1.006, n=34 | 1
  Week 32, USG, 1.007, n=34 | 1
  Week 32, USG, 1.01, n=34 | 4
  Week 32, USG, 1.011, n=34 | 1
  Week 32, USG, 1.012, n=34 | 1
  Week 32, USG, 1.014, n=34 | 1
  Week 32, USG, 1.015, n=34 | 4
  Week 32, USG, 1.016, n=34 | 3
  Week 32, USG, 1.018, n=34 | 2
  Week 32, USG, 1.019, n=34 | 1
  Week 32, USG, 1.02, n=34 | 6
  Week 32, USG, 1.021, n=34 | 3
  Week 32, USG, 1.022, n=34 | 3
  Week 32, USG, 1.024, n=34 | 1
  Week 32, UU, 1+, n=34 | 3
  Week 32, UU, 0.1, n=34 | 2
  Week 32, UU, 1, n=34 | 7
  Week 32, UU, 3, n=34 | 1
  Week 32, UU, 4, n=34 | 1
  Week 32, UU, 8, n=34 | 1
  Week 32, UU, Neg, n=34 | 1
  Week 32, UU, trace, n=34 | 12
  Week 32, UU, normal, n=34 | 6
  Week 36, UB, 1+, n=34 | 1
  Week 36, UB, (-), n=34 | 1
  Week 36, UB, Neg, n=34 | 32
  Week 36, UOB, 2+, n=34 | 2
  Week 36, UOB, (-), n=34 | 1
  Week 36, UOB, Neg, n=34 | 31
  Week 36, UG, (-), n=34 | 1
  Week 36, UG, Neg, n=34 | 33
  Week 36, UK, 1+, n=34 | 1
  Week 36, UK, (-), n=34 | 1
  Week 36, UK, Neg, n=34 | 32
  Week 36, pH, 5, n=34 | 1
  Week 36, pH, 5.5, n=34 | 3
  Week 36, pH, 6, n=34 | 9
  Week 36, pH, 6.5, n=34 | 7
  Week 36, pH, 7, n=34 | 10
  Week 36, pH, 7.5, n=34 | 4
  Week 36, UP, 1+, n=34 | 1
  Week 36, UP, (-), n=34 | 1
  Week 36, UP, Neg, n=34 | 30
  Week 36, UP, trace, n=34 | 2
  Week 36, USG, 1.005, n=34 | 2
  Week 36, USG, 1.007, n=34 | 1
  Week 36, USG, 1.008, n=34 | 2
  Week 36, USG, 1.009, n=34 | 2
  Week 36, USG, 1.01, n=34 | 2
  Week 36, USG, 1.011, n=34 | 1
  Week 36, USG, 1.012, n=34 | 2
  Week 36, USG, 1.013, n=34 | 3
  Week 36, USG, 1.015, n=34 | 3
  Week 36, USG, 1.016, n=34 | 2
  Week 36, USG, 1.018, n=34 | 2
  Week 36, USG, 1.02, n=34 | 4
  Week 36, USG, 1.021, n=34 | 4
  Week 36, USG, 1.023, n=34 | 1
  Week 36, USG, 1.024, n=34 | 1
  Week 36, USG, 1.03, n=34 | 1
  Week 36, USG, <=1.005, n=34 | 1
  Week 36, UU, 1+, n=34 | 2
  Week 36, UU, 0.1, n=34 | 3
  Week 36, UU, 1, n=34 | 7
  Week 36, UU, 2, n=34 | 1
  Week 36, UU, 3, n=34 | 1
  Week 36, UU, 4, n=34 | 1
  Week 36, UU, Neg, n=34 | 1
  Week 36, UU, trace, n=34 | 14
  Week 36, UU, normal, n=34 | 4
  Week 40, UB, (-), n=33 | 1
  Week 40, UB, Neg, n=33 | 32
  Week 40, UOB, 2+, n=33 | 1
  Week 40, UOB, 3+, n=33 | 1
  Week 40, UOB, (-), n=33 | 1
  Week 40, UOB, Neg, n=33 | 30
  Week 40, UG, (-), n=33 | 1
  Week 40, UG, Neg, n=33 | 32
  Week 40, UK, (-), n=33 | 1
  Week 40, UK, Neg, n=33 | 31
  Week 40, UK, trace, n=33 | 1
  Week 40, pH, 5.5, n=33 | 4
  Week 40, pH, 6, n=33 | 9
  Week 40, pH, 6.5, n=33 | 6
  Week 40, pH, 7, n=33 | 10
  Week 40, pH, 7.5, n=33 | 4
  Week 40, UP, (-), n=33 | 1
  Week 40, UP, Neg, n=33 | 30
  Week 40, UP, trace, n=33 | 2
  Week 40, USG, 1.003, n=33 | 1
  Week 40, USG, 1.004, n=33 | 1
  Week 40, USG, 1.005, n=33 | 2
  Week 40, USG, 1.006, n=33 | 1
  Week 40, USG, 1.007, n=33 | 2
  Week 40, USG, 1.01, n=33 | 2
  Week 40, USG, 1.011, n=33 | 1
  Week 40, USG, 1.012, n=33 | 3
  Week 40, USG, 1.013, n=33 | 3
  Week 40, USG, 1.014, n=33 | 1
  Week 40, USG, 1.015, n=33 | 1
  Week 40, USG, 1.016, n=33 | 3
  Week 40, USG, 1.018, n=33 | 1
  Week 40, USG, 1.019, n=33 | 2
  Week 40, USG, 1.02, n=33 | 4
  Week 40, USG, 1.022, n=33 | 1
  Week 40, USG, 1.023, n=33 | 2
  Week 40, USG, 1.024, n=33 | 1
  Week 40, USG, 1.025, n=33 | 1
  Week 40, UU, 1+, n=33 | 1
  Week 40, UU, 0.1, n=33 | 3
  Week 40, UU, 1, n=33 | 6
  Week 40, UU, 2, n=33 | 1
  Week 40, UU, 3, n=33 | 1
  Week 40, UU, 4, n=33 | 1
  Week 40, UU, Neg, n=33 | 1
  Week 40, UU, trace, n=33 | 13
  Week 40, UU, normal, n=33 | 6
  Week 44, UB, (-), n=31 | 1
  Week 44, UB, Neg, n=31 | 30
  Week 44, UOB, 2+, n=31 | 2
  Week 44, UOB, (-), n=31 | 1
  Week 44, UOB, Neg, n=31 | 28
  Week 44, UG, (-), n=31 | 1
  Week 44, UG, 0.1, n=31 | 1
  Week 44, UG, Neg, n=31 | 29
  Week 44, UK, (-), n=31 | 1
  Week 44, UK, Neg, n=31 | 29
  Week 44, UK, trace, n=31 | 1
  Week 44, pH, 5.5, n=31 | 3
  Week 44, pH, 6, n=31 | 12
  Week 44, pH, 6.5, n=31 | 8
  Week 44, pH, 7, n=31 | 6
  Week 44, pH, 7.5, n=31 | 2
  Week 44, UP, (-), n=31 | 1
  Week 44, UP, Neg, n=31 | 27
  Week 44, UP, trace, n=31 | 3
  Week 44, USG, 1.005, n=31 | 3
  Week 44, USG, 1.007, n=31 | 2
  Week 44, USG, 1.008, n=31 | 2
  Week 44, USG, 1.01, n=31 | 3
  Week 44, USG, 1.011, n=31 | 3
  Week 44, USG, 1.012, n=31 | 1
  Week 44, USG, 1.015, n=31 | 1
  Week 44, USG, 1.016, n=31 | 1
  Week 44, USG, 1.017, n=31 | 3
  Week 44, USG, 1.018, n=31 | 1
  Week 44, USG, 1.019, n=31 | 1
  Week 44, USG, 1.02, n=31 | 2
  Week 44, USG, 1.021, n=31 | 2
  Week 44, USG, 1.022, n=31 | 1
  Week 44, USG, 1.024, n=31 | 1
  Week 44, USG, 1.025, n=31 | 2
  Week 44, USG, 1.027, n=31 | 1
  Week 44, USG, 1.03, n=31 | 1
  Week 44, UU, 1+, n=31 | 3
  Week 44, UU, 2+, n=31 | 1
  Week 44, UU, 0.1, n=31 | 3
  Week 44, UU, 1, n=31 | 7
  Week 44, UU, 2, n=31 | 1
  Week 44, UU, 4, n=31 | 1
  Week 44, UU, Neg, n=31 | 1
  Week 44, UU, trace, n=31 | 11
  Week 44, UU, normal, n=31 | 3
  Week 48, UB, (-), n=31 | 1
  Week 48, UB, Neg, n=31 | 30
  Week 48, UOB, 3+, n=31 | 1
  Week 48, UOB, (-), n=31 | 1
  Week 48, UOB, Neg, n=31 | 29
  Week 48, UG, (-), n=31 | 1
  Week 48, UG, Neg, n=31 | 30
  Week 48, UK, (-), n=31 | 1
  Week 48, UK, Neg, n=31 | 30
  Week 48, pH, 5.5, n=31 | 4
  Week 48, pH, 6, n=31 | 6
  Week 48, pH, 6.5, n=31 | 14
  Week 48, pH, 7, n=31 | 6
  Week 48, pH, 8, n=31 | 1
  Week 48, UP, (-), n=31 | 1
  Week 48, UP, 10, n=31 | 1
  Week 48, UP, Neg, n=31 | 26
  Week 48, UP, trace, n=31 | 3
  Week 48, USG, 1.005, n=31 | 1
  Week 48, USG, 1.007, n=31 | 1
  Week 48, USG, 1.009, n=31 | 2
  Week 48, USG, 1.01, n=31 | 3
  Week 48, USG, 1.011, n=31 | 2
  Week 48, USG, 1.012, n=31 | 1
  Week 48, USG, 1.013, n=31 | 1
  Week 48, USG, 1.014, n=31 | 1
  Week 48, USG, 1.015, n=31 | 4
  Week 48, USG, 1.016, n=31 | 1
  Week 48, USG, 1.017, n=31 | 1
  Week 48, USG, 1.018, n=31 | 4
  Week 48, USG, 1.019, n=31 | 3
  Week 48, USG, 1.02, n=31 | 2
  Week 48, USG, 1.025, n=31 | 2
  Week 48, USG, 1.027, n=31 | 1
  Week 48, USG, 1.03, n=31 | 1
  Week 48, UU, 1+, n=31 | 2
  Week 48, UU, 0.1, n=31 | 4
  Week 48, UU, 1, n=31 | 3
  Week 48, UU, 2, n=31 | 2
  Week 48, UU, 3, n=31 | 1
  Week 48, UU, Neg, n=31 | 1
  Week 48, UU, trace, n=31 | 14
  Week 48, UU, normal, n=31 | 4
  Withdrawal, UB, 1+, n=10 | 1
  Withdrawal, UB, (-), n=10 | 1
  Withdrawal, UB, Neg, n=10 | 8
  Withdrawal, UOB, 1+, n=10 | 1
  Withdrawal, UOB, (-), n=10 | 2
  Withdrawal, UOB, Neg, n=10 | 7
  Withdrawal, UG, (-), n=10 | 2
  Withdrawal, UG, Neg, n=10 | 8
  Withdrawal, UK, (-), n=10 | 2
  Withdrawal, UK, Neg, n=10 | 8
  Withdrawal, pH, 5, n=10 | 1
  Withdrawal, pH, 6, n=10 | 5
  Withdrawal, pH, 6.5, n=10 | 2
  Withdrawal, pH, 7, n=10 | 2
  Withdrawal, UP, Neg, n=10 | 5
  Withdrawal, UP, trace, n=10 | 5
  Withdrawal, USG, 1.002, n=10 | 1
  Withdrawal, USG, 1.009, n=10 | 1
  Withdrawal, USG, 1.01, n=10 | 1
  Withdrawal, USG, 1.017, n=10 | 1
  Withdrawal, USG, 1.018, n=10 | 1
  Withdrawal, USG, 1.019, n=10 | 2
  Withdrawal, USG, 1.021, n=10 | 1
  Withdrawal, USG, 1.023, n=10 | 1
  Withdrawal, USG, 1.025, n=10 | 1
  Withdrawal, UU, 1+, n=10 | 2
  Withdrawal, UU, 1, n=10 | 1
  Withdrawal, UU, Neg, n=10 | 1
  Withdrawal, UU, trace, n=10 | 3
  Withdrawal, UU, normal, n=10 | 3

52. Secondary Outcome: Number of Participants With the Indicated Urinalysis Parameters Tested by Dipstick at the Indicated Time Points During Follow-up Period After Part 2
Description: as for outcome 51
Time Frame: FU Baseline and FU Week 24
Population: SP2 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2
Number analyzed (Participants) | 37
Participants
  FU Baseline, UB, (-) | 3
  FU Baseline, UB, Neg. | 34
  FU Baseline, UOB, 1+ | 1
  FU Baseline, UOB, 3+ | 1
  FU Baseline, UOB, (-) | 3
  FU Baseline, UOB, Neg. | 32
  FU Baseline, UG, (-) | 3
  FU Baseline, UG, Neg | 34
  FU Baseline, UK, (-) | 3
  FU Baseline, UK, Neg. | 34
  FU Baseline, pH, 5 | 1
  FU Baseline, pH, 5.5 | 4
  FU Baseline, pH, 6 | 10
  FU Baseline, pH, 6.5 | 13
  FU Baseline, pH, 7 | 8
  FU Baseline, pH, 8 | 1
  FU Baseline, UP, (-) | 1
  FU Baseline, UP, 10 | 1
  FU Baseline, UP, Neg | 27
  FU Baseline, UP, trace | 8
  FU Baseline, USG, 1.002 | 1
  FU Baseline, USG, 1.005 | 1
  FU Baseline, USG, 1.007 | 1
  FU Baseline, USG, 1.009 | 2
  FU Baseline, USG, 1.01 | 2
  FU Baseline, USG, 1.011 | 2
  FU Baseline, USG, 1.012 | 1
  FU Baseline, USG, 1.013 | 1
  FU Baseline, USG, 1.014 | 1
  FU Baseline, USG, 1.015 | 4
  FU Baseline, USG, 1.016 | 1
  FU Baseline, USG, 1.017 | 2
  FU Baseline, USG, 1.018 | 4
  FU Baseline, USG, 1.019 | 5
  FU Baseline, USG, 1.02 | 2
  FU Baseline, USG, 1.021 | 1
  FU Baseline, USG, 1.024 | 1
  FU Baseline, USG, 1.025 | 3
  FU Baseline, USG, 1.027 | 1
  FU Baseline, USG, 1.03 | 1
  FU Baseline, UU, 1+ | 4
  FU Baseline, UU, 0.1 | 3
  FU Baseline, UU, 1 | 3
  FU Baseline, UU, 2 | 1
  FU Baseline, UU, 3 | 1
  FU Baseline, UU, Neg | 2
  FU Baseline, UU, trace | 17
  FU Baseline, UU, normal | 6
  FU Week 24, UB, (-) | 2
  FU Week 24, UB, Neg. | 35
  FU Week 24, UOB, 1+ | 3
  FU Week 24, UOB, 3+ | 1
  FU Week 24, UOB, (-) | 2
  FU Week 24, UOB, Neg. | 26
  FU Week 24, UOB, Trace | 5
  FU Week 24, UG, 1+ | 1
  FU Week 24, UG, (-) | 2
  FU Week 24, UG, 0.2 | 1
  FUWeek 24, UG, Neg | 33
  FU Week 24, UK, (-) | 2
  FU Week 24, UK, Neg. | 34
  FU Week 24, UK, Trace. | 1
  FU Week 24, pH, 5 | 4
  FU Week 24, pH, 5.5 | 9
  FU Week 24, pH, 6 | 7
  FU Week 24, pH, 6.5 | 10
  FU Week 24, pH, 7 | 3
  FU Week 24, pH, 7.5 | 4
  FU Week 24, UP, (-) | 2
  FU Week 24, UP, Neg | 32
  FU Week 24, UP, Trace | 3
  FU Week 24, USG, 1.004 | 1
  FU Week 24, USG, 1.005 | 2
  FU Week 24, USG, 1.008 | 2
  FU Week 24, USG, 1.01 | 5
  FU Week 24, USG, 1.011 | 4
  FU Week 24, USG, 1.012 | 1
  FU Week 24, USG, 1.013 | 2
  FU Week 24, USG, 1.015 | 3
  FU Week 24, USG, 1.016 | 2
  FU Week 24, USG, 1.017 | 4
  FU Week 24, USG, 1.018 | 1
  FU Week 24, USG, 1.019 | 1
  FU Week 24, USG, 1.02 | 2
  FU Week 24, USG, 1.021 | 2
  FU Week 24, USG, 1.022 | 2
  FU Week 24, USG, 1.023 | 1
  FU Week 24, USG, 1.024 | 1
  FU Week 24, USG, 1.025 | 1
  FU Week 24, UU, 0.1 | 5
  FU Week 24, UU, 1 | 2
  FU Week 24, UU, 4 | 1
  FU Week 24, UU, <1.0 | 1
  FU Week 24, UU, Neg | 2
  FU Week 24, UU, Trace | 18
  FUWeek 24, UU, normal | 8

53. Secondary Outcome: Number of Participants Assessed as Abnormal (Clinically Significant [CS] and Not Clinically Significant [NCS]) for 12-lead Electrocardiogram (ECG) at the Indicated Time Points
Description: The number of participants with an ECG status of normal, abnormal, CS, or NCS, as determined by the Investigator, was reported. Normal= all ECG parameters within accepted normal ranges. Abnormal= ECG findings outside of normal ranges. CS= ECG with a CS abnormality that meets exclusion criteria. NCS= ECG with an abnormality not CS or meeting exclusion criteria, per Investigator, based on reasonable standards of clinical judgment.
Time Frame: Screening, Antiviral Baseline, Week 12, 24, 36, 48, Withdrawal
Population: SP1 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag Dose Escalation: Part 1
Number analyzed (Participants) | 45
Participants
  Screening, normal, n=45 | 31
  Screening, abnormal-NCS, n=45 | 14
  Screening, abnormal-CS, n=45 | 0
  Antiviral Baseline, normal, n=41 | 26
  Antiviral Baseline, abnormal-NCS, n=41 | 14
  Antiviral Baseline, abnormal-CS, n=41 | 1
  Part 2, week 12, normal, n=36 | 29
  Part 2, week 12, abnormal-NCS, n=36 | 7
  Part 2, week 12, abnormal-CS, n=36 | 0
  Part 2, week 24, normal, n=36 | 29
  Part 2, week 24, abnormal-NCS, n=36 | 7
  Part 2, week 24, abnormal-CS, n=36 | 0
  Part 2, week 36, normal, n=34 | 24
  Part 2, week 36, abnormal-NCS, n=34 | 10
  Part 2, week 36, abnormal-CS, n=34 | 0
  Part 2, week 48, normal, n=31 | 19
  Part 2, week 48, abnormal-NCS, n=31 | 12
  Part 2, week 48, abnormal-CS, n=31 | 0
  Withdrawal, normal, n=14 | 10
  Withdrawal, abnormal-NCS, n=14 | 4
  Withdrawal, abnormal-CS, n=14 | 0
  Worst ECG post Baseline, normal, n=41 | 24
  Worst ECG post Baseline, abnormal-NCS, n=41 | 17
  Worst ECG post Baseline, abnormal-CS, n=41 | 0

54. Secondary Outcome: Number of Participants Assessed as Abnormal (Clinically Significant [CS] and Not Clinically Significant [NCS]) for 12-lead Electrocardiogram (ECG) During Follow-up After Part 2
Description: as for outcome 53
Time Frame: FU Baseline and FU Week 24
Population: SP2 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2
Number analyzed (Participants) | 37
Participants
  FU Baseline, normal | 24
  FU Baseline, abnormal-NCS | 13
  FU Baseline, abnormal-CS | 0
  FU Week 24, normal | 31
  FU Week 24, abnormal-NCS | 6
  FU Week 24, abnormal-CS | 0

55. Secondary Outcome: Number of Participants With Abdominal Ultrasound With Doppler at the Indicated Time Points
Description: Abdominal ultrasound with doppler were taken at Baseline, Week 24, Week 48, withdrawal (WD)/completion (comp). Questions were asked to assess masses suspicious for hepatocellular carcinoma (HCC), ascites, portal vein thrombosis detected, possiblility to measure spleen breadth, and other clinically significant findings (OCSF).
Time Frame: Baseline; Week 24, Week 48, Withdrawal/Completion
Population: SP1 Population. Only those participants available at the specified time points were analyzed (n=X).
Measure: Number; unit: Participants
Arm/Group | Eltrombopag Dose Escalation: Part 1
Number analyzed (Participants) | 45
Participants
  Baseline, masses suspicious for HCC detected, n=45 | 0
  Baseline, ascites detected, n=45 | 0
  Baseline, portal vein thrombosis detected, n=45 | 0
  Baseline, measureable spleen breadth, n=45 | 43
  Baseline, OCSF, n=45 | 8
  Week 24, masses suspicious for HCC detected, n=36 | 1
  Week 24, ascites detected, n=36 | 1
  Week 24, portal vein thrombosis detected, n=36 | 0
  Week 24, measureable spleen breadth, n=36 | 34
  Week 24, OCSF, n=36 | 4
  Week 48, masses suspicious for HCC detected, n=29 | 0
  Week 48, ascites detected, n=29 | 1
  Week 48, portal vein thrombosis detected, n=29 | 0
  Week 48, measureable spleen breadth, n=29 | 29
  Week 48, OCSF, n=29 | 3
  WD/comp, masses suspicious for HCC detected, n=37 | 2
  WD/comp, ascites detected, n=37 | 2
  WD/comp, portal vein thrombosis detected, n=37 | 0
  WD/comp, measureable spleen breadth, n=37 | 37
  WD/comp, OCSF, n=37 | 6

56. Secondary Outcome: Number of Participants With Abdominal Ultrasound With Doppler During Follow-up Period After Part 2
Description: Abdominal ultrasound with doppler were taken during Follow-up Period after Part 2 at FU Week 24. Questions were asked to assess masses suspicious for hepatocellular carcinoma (HCC), ascites, portal vein thrombosis detected, possiblility to measure spleen breadth, and other clinically significant findings (OCSF).
Time Frame: FU Week 24
Population: SP2 Population.
Measure: Number; unit: Participants
Arm/Group | Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2
Number analyzed (Participants) | 36
Participants
  FU Week 24, masses suspicious for HCC detected, | 1
  FU Week 24, ascites detected | 1
  FU Week 24, portal vein thrombosis detected | 0
  FU Week 24, measureable spleen breadth | 36
  FU Week 24, OCSF | 4

57. Secondary Outcome: Spleen Measurements as Assessed by Abdominal Ultrasound With Doppler in the Study
Description: Abdominal ultrasound with doppler were taken at Baseline, Week 24, Week 48, WD/comp. Questions were asked to assess masses suspicious for HCC, ascites, portal vein thrombosis detected, possiblility to measure spleen breadth, and OCSF. Spleen measurements included spleen length and spleen width (breadth).
Time Frame: Baseline; Week 24, Week 48, Withdrawal/Completion
Population: SP1 Population. Only those participants available at the specified time points were analyzed (n=X).
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Eltrombopag Dose Escalation: Part 1
Number analyzed (Participants) | 45
Centimeters (cm)
  Baseline, spleen length, n=45 | 11.5 (2.63)
  Baseline, spleen width (breadth), n=43 | 4.7 (1.25)
  Week 24, spleen length, n=36 | 11.5 (2.34)
  Week 24, spleen width (breadth), n=34 | 4.9 (1.21)
  Week 48, spleen length, n=29 | 11.6 (2.27)
  Week 48, spleen width (breadth), n=29 | 4.5 (0.87)
  WD/comp, spleen length, n=37 | 11.7 (2.67)
  WD/comp, spleen width (breadth), n=37 | 4.5 (0.93)

58. Secondary Outcome: Spleen Measurements as Assessed by Abdominal Ultrasound With Doppler During Follow-up Period After Part 2
Description: Abdominal ultrasound with doppler were taken during Follow-up Period after Part 2 at FU Week 24. Questions were asked to assess masses suspicious for HCC, ascites, portal vein thrombosis detected, possiblility to measure spleen breadth, and OCSF. Spleen measurements included spleen length and spleen width (breadth).
Time Frame: FU Week 24
Population: SP2 Population.
Measure: Mean (Standard Deviation); unit: Cm
Arm/Group | Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2
Number analyzed (Participants) | 36
Cm
  FU Week 24, spleen length | 11.0 (2.61)
  FU Week 24, spleen width (breadth) | 4.4 (1.32)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from start of study medication until follow-up visit (up to a maximun of 81 weeks).
Description: SAEs and non-serious AEs are reported for members of the Safety Population, comprised of all participants enrolled in the Pre-Antiviral Treatment Period and Antivital Treatment Period, who received at least one dose of eltrombopag.
Arm/Group | Eltrombopag Dose Escalation: Part 1 | Eltrombopag + Antiviral Therapy: Part 2 | Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2
Serious Adverse Events (participants affected / at risk) | 0/45 | 3/41 | 4/41
Other Adverse Events (participants affected / at risk) | 0/45 | 41/41 | 6/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag Dose Escalation: Part 1 (N=45) | Eltrombopag + Antiviral Therapy: Part 2 (N=41) | Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2 (N=41)
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Myeloblast percentage increased (Investigations) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag Dose Escalation: Part 1 (N=45) | Eltrombopag + Antiviral Therapy: Part 2 (N=41) | Eltrombopag + Antiviral Therapy: Follow-up Period After Part 2 (N=41)
Anaemia (Blood and lymphatic system disorders) | 0 | 22 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 17 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 8 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 7 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 16 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 14 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 13 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 7 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 12 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 6 | 0
Nausea (Gastrointestinal disorders) | 0 | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 5 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 4 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 0
Dental caries (Gastrointestinal disorders) | 0 | 3 | 0
Toothache (Gastrointestinal disorders) | 0 | 3 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0
Pyrexia (General disorders) | 0 | 24 | 0
Malaise (General disorders) | 0 | 11 | 0
Fatigue (Gastrointestinal disorders) | 0 | 4 | 0
Injection site erythema (General disorders) | 0 | 4 | 0
Injection site pruritus (General disorders) | 0 | 4 | 0
Injection site reaction (General disorders) | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 9 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 7 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0
Headache (Nervous system disorders) | 0 | 13 | 0
Dysgeusia (Nervous system disorders) | 0 | 5 | 0
Dizziness (Nervous system disorders) | 0 | 4 | 0
Retinal haemorrhage (Eye disorders) | 0 | 7 | 0
Retinopathy (Eye disorders) | 0 | 6 | 0
Retinal exudates (Eye disorders) | 0 | 5 | 0
White blood cell count decreased (Investigations) | 0 | 7 | 0
Weight decreased (Investigations) | 0 | 6 | 0
Neutrophil count decreased (Investigations) | 0 | 5 | 0
Haemoglobin decreased (Investigations) | 0 | 4 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 9 | 0
Cystitis (Infections and infestations) | 0 | 4 | 0
Enteritis infectious (Infections and infestations) | 0 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 9 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0
Insomnia (Psychiatric disorders) | 0 | 6 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.